CLINICAL TRIAL: NCT02712983
Title: A Randomized, Blinded, Parallel Group, Multi-center Dose-finding Study, to Assess the Efficacy, Safety and Tolerability of Different Doses of Tobramycin Inhalation Powder in Patients With Non-Cystic Fibrosis Bronchiectasis and Pulmonary P. Aeruginosa Infection
Brief Title: Dose-finding Study to Assess the Efficacy, Safety and Tolerability of Tobramycin Inhalation Powder in Patients With Non-Cystic Fibrosis Bronchiectasis and Pulmonary P. Aeruginosa Infection
Acronym: iBEST-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: Queen's University, Belfast (Other); University Hospital, Antwerp (Other); University of Milan (Other); Fundacion Clinic per a la Recerca Biomédica (Other); Erasmus Medical Center (Other); Papworth Hospital NHS Foundation Trust (Other Government); Royal Brompton & Harefield NHS Foundation Trust (Other); University of Dundee (Other); University of Edinburgh (Other)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CTBM100G2202; 2015-003040-39 (EudraCT Number)
Record Dates: First submitted 2016-02-05; First posted 2016-03-18 (Estimated); Results first posted 2020-08-14 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Non-cystic Fibrosis Bronchiectasis
Keywords: Inhaled tobramycin; tobramycin inhalation powder; bronchiectasis; pulmonary Pseudomonas aeruginosa infection; dose-finding study
MeSH Terms: conditions — Bronchiectasis | interventions — Lysine Acetyltransferase 5

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Cohort A (3 capsules o.d.): TIP (Experimental): Cohort A (3 capsules o.d.): Tobramycin inhalation powder (TIP)
  Interventions: Drug: TIP
- Cohort A (3 capsules o.d.): TIP/PBO (Experimental): Cohort A (3 capsules o.d.): Tobramycin inhalation powder (TIP) and inhaled placebo (PBO) cyclical
  Interventions: Drug: TIP and placebo
- Cohort A (3 capsules o.d.): PBO (Placebo Comparator): Cohort A (3 capsules o.d.): Inhaled placebo (PBO)
  Interventions: Drug: Placebo
- Cohort B (5 capsules o.d.): TIP (Experimental): Cohort B (5 capsules o.d.): Tobramycin inhalation powder (TIP)
  Interventions: Drug: TIP
- Cohort B (5 capsules o.d.): TIP/PBO (Experimental): Cohort B (5 capsules o.d.): Tobramycin inhalation powder (TIP) and inhaled placebo (PBO) cyclical
  Interventions: Drug: TIP and placebo
- Cohort B (5 capsules o.d.): PBO (Placebo Comparator): Cohort B (5 capsules o.d.): inhaled placebo (PBO)
  Interventions: Drug: Placebo
- Cohort C (4 capsules b.i.d.): TIP (Experimental): Cohort C (4 capsules b.i.d.): Tobramycin inhalation powder (TIP)
  Interventions: Drug: TIP
- Cohort C (4 capsules b.i.d.): TIP/PBO (Experimental): Cohort C (4 capsules b.i.d.): Tobramycin inhalation powder (TIP) and inhaled placebo (PBO) cyclical
  Interventions: Drug: TIP and placebo
- Cohort C (4 capsules b.i.d.): PBO (Placebo Comparator): Cohort C (4 capsules b.i.d.): inhaled placebo (PBO)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TIP — TIP dose regimen
  Arms: Cohort A (3 capsules o.d.): TIP; Cohort B (5 capsules o.d.): TIP; Cohort C (4 capsules b.i.d.): TIP
Drug: TIP and placebo — TIP and inhaled placebo dose regimen
  Arms: Cohort A (3 capsules o.d.): TIP/PBO; Cohort B (5 capsules o.d.): TIP/PBO; Cohort C (4 capsules b.i.d.): TIP/PBO
Drug: Placebo — Inhaled placebo dose regimen
  Arms: Cohort A (3 capsules o.d.): PBO; Cohort B (5 capsules o.d.): PBO; Cohort C (4 capsules b.i.d.): PBO

SUMMARY:
The purpose of this study was to support the selection of a safe and tolerable tobramycin inhalation powder (TIP) dose, and regimen that exhibits effective bacterial reduction of P. aeruginosa in non-cystic fibrosis bronchiectasis (BE) patients with P. aeruginosa colonization.

DETAILED DESCRIPTION:
This was a blinded, randomized, dose and regimen finding trial utilizing a three treatment cohort design where active TIP and TIP/Placebo cyclical (3 capsules o.d [Cohort A], 5 capsules o.d. [Cohort B] or 4 capsules b.i.d. [Cohort C]) versus Placebo were administered for a total of 112 days.

Novartis decided to close the recruitment of new subjects into this study earlier than scheduled. Subjects who had a signed informed consent form and entered screening by 10-Sep-2018 still participated in the study. The latest possible randomization was on 08-Oct-2018. All subjects enrolled in the study (107 enrolled subjects out of 180 planned) continued as planned through to their last scheduled visit. The early recruitment halt of the study was not due to safety or lack of efficacy.

ELIGIBILITY:
Key Inclusion Criteria:

* Written informed consent must be obtained before any assessment is performed.
* Male and female patients of ≥ 18 years of age at screening (Visit 1).
* Proven diagnosis of non-CF BE as documented by computed tomography or high-resolution computed tomography
* At least 2 or more exacerbations treated with oral antibiotics OR 1 or more exacerbation requiring intravenous antibiotic treatment within 12 months prior to screening.
* FEV1 ≥ 30% predicted at screening (Visit 1).
* P. aeruginosa, must be documented in a respiratory sample at least 1 time within 12 months and also present in the expectorated sputum culture at Visit 1.

Key Exclusion Criteria:

* Patients with a history of cystic fibrosis.
* Patients with a primary diagnosis of bronchial asthma.
* Patients with a primary diagnosis of COPD associated with at least a 20 pack year smoking history.
* Any significant medical condition that is either recently diagnosed or was not stable during the last 3 months, other than pulmonary exacerbations, and that in the opinion of the investigator makes participation in the trial against the patients' best interests.
* Clinically significant (in the opinion of the investigator) hearing loss that interferes with patients' daily activities (such as normal conversations) or chronic tinnitus. Patients with a past history of clinically significant hearing loss in the opinion of the investigator may be eligible only if their hearing threshold at screening audiometry is 25dB or lower at frequencies 0.5-4 kHz. The use of a hearing device is reflective of a clinically significant hearing loss; hence patients using hearing aids at screening are not eligible.
* Patients with active pulmonary tuberculosis.
* Patients currently receiving treatment for nontuberculous mycobacterial (NTM) pulmonary disease.
* Patients who are regularly receiving inhaled anti-pseudomonal antibiotic (during the study inhaled anti-pseudomonal antibiotics are not allowed other than the study drug).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2017-02-08 (Actual); Primary Completion 2019-03-20 (Actual); Study Completion 2019-03-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharma, Study Director — Novartis Pharmaceuticals
Locations (32):
- Belgium (2):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Leuven
- France (4):
  - Novartis Investigative Site, Nice, Cedex1
  - Novartis Investigative Site, Montpellier, Herault
  - Novartis Investigative Site, Grenoble
  - Novartis Investigative Site, Toulouse
- Germany (5):
  - Novartis Investigative Site, Essen, North Rhine-Westphalia
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Leipzig
- Italy (6):
  - Novartis Investigative Site, Monza, MB
  - Novartis Investigative Site, Pisa, PI
  - Novartis Investigative Site, Pordenone, PN
  - Novartis Investigative Site, Milan
  - Novartis Investigative Site, Pavia
  - Novartis Investigative Site, Scafati
- Spain (6):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Valencia, Comunitat Valencia
  - Novartis Investigative Site, Baracaldo - Vizcaya
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Valencia
  - Novartis Investigative Site, Valladolid
- United Kingdom (9):
  - Novartis Investigative Site, Cambridge, Cambridgeshire
  - Novartis Investigative Site, Dundee, Perthshire
  - Novartis Investigative Site, Birmingham
  - Novartis Investigative Site, Edinburgh
  - Novartis Investigative Site, Lancaster
  - Novartis Investigative Site, Leeds
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Newcastle upon Tyne
  - Novartis Investigative Site, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Loebinger MR, Polverino E, Chalmers JD, Tiddens HAWM, Goossens H, Tunney M, Ringshausen FC, Hill AT, Pathan R, Angyalosi G, Blasi F, Elborn SJ, Haworth CS; iBEST-1 Trial Team. Efficacy and safety of TOBI Podhaler in Pseudomonas aeruginosa-infected bronchiectasis patients: iBEST study. Eur Respir J. 2021 Jan 5;57(1):2001451. doi: 10.1183/13993003.01451-2020. Print 2021 Jan. PMID 32855225
- [Derived] Loebinger MR, Polverino E, Blasi F, Elborn SJ, Chalmers JD, Tiddens HA, Goossens H, Tunney M, Zhou W, Angyalosi G, Hill AT, Haworth CS; iBEST-1 Trial Team. Efficacy and safety of tobramycin inhalation powder in bronchiectasis patients with P. aeruginosa infection: Design of a dose-finding study (iBEST-1). Pulm Pharmacol Ther. 2019 Oct;58:101834. doi: 10.1016/j.pupt.2019.101834. Epub 2019 Aug 18. PMID 31433997

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 107 subjects were enrolled in the trial from 6 countries (Belgium [2 sites], France [4 sites], Germany [5 sites], Italy [6 sites], Spain [8 sites] and United Kingdom [9 sites]).
Pre-assignment Details: This study planned to recruit approximately 180 subjects to one of the 3 cohorts in a ratio of 1:1:1. The subjects within each cohort were randomized to blinded TIP or placebo with the following randomization scheme: TIP:TIP/Placebo cyclical:Placebo, in a 2:2:1 ratio.
Period: Treatment Phase
Arm/Group | Cohort A (3 Capsules o.d.): TIP | Cohort A (3 Capsules o.d.): TIP/PBO | Cohort A (3 Capsules o.d.): PBO | Cohort B (5 Capsules o.d.): TIP | Cohort B (5 Capsules o.d.): TIP/PBO | Cohort B (5 Capsules o.d.): PBO | Cohort C (4 Capsules b.i.d.): TIP | Cohort C (4 Capsules b.i.d.): TIP/PBO | Cohort C (4 Capsules b.i.d.): PBO
Started (All randomized patients (Full Analysis Set and Safety Set)) | 14 | 13 | 7 | 15 | 14 | 7 | 15 | 15 | 7
Pharmacokinetic Analysis Set | 14 | 13 | 0 | 15 | 14 | 0 | 15 | 14 | 0
Completed | 9 | 12 | 6 | 7 | 10 | 7 | 6 | 6 | 5
Not Completed | 5 | 1 | 1 | 8 | 4 | 0 | 9 | 9 | 2
Not completed — Adverse Event | 3 | 1 | 1 | 4 | 3 | 0 | 6 | 6 | 1
Not completed — Protocol Deviation | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0
Not completed — Technical Problems | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Subject Decision | 2 | 0 | 0 | 2 | 1 | 0 | 1 | 2 | 0
Period: Post-Treatment Efficacy Follow-Up Phase
Arm/Group | Cohort A (3 Capsules o.d.): TIP | Cohort A (3 Capsules o.d.): TIP/PBO | Cohort A (3 Capsules o.d.): PBO | Cohort B (5 Capsules o.d.): TIP | Cohort B (5 Capsules o.d.): TIP/PBO | Cohort B (5 Capsules o.d.): PBO | Cohort C (4 Capsules b.i.d.): TIP | Cohort C (4 Capsules b.i.d.): TIP/PBO | Cohort C (4 Capsules b.i.d.): PBO
Started (All patients who discontinued treatment and entered Post-Treatment Efficacy Follow-Up Phase) | 0 (All patients who entered Post-Treatment Efficacy Fup Phase) | 1 (All patients who entered Post-Treatment Efficacy Fup Phase) | 0 (All patients who entered Post-Treatment Efficacy Fup Phase) | 1 (All patients who entered Post-Treatment Efficacy Fup Phase) | 2 (All patients who entered Post-Treatment Efficacy Fup Phase) | 1 (All patients who entered Post-Treatment Efficacy Fup Phase) | 2 (All patients who entered Post-Treatment Efficacy Fup Phase) | 3 (All patients who entered Post-Treatment Efficacy Fup Phase) | 0 (All patients who entered Post-Treatment Efficacy Fup Phase)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 1 | 0 | 1 | 2 | 1 | 2 | 3 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Subject Decision | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A (3 Capsules o.d.): TIP | Cohort A (3 Capsules o.d.): TIP/PBO | Cohort A (3 Capsules o.d.): PBO | Cohort B (5 Capsules o.d.): TIP | Cohort B (5 Capsules o.d.): TIP/PBO | Cohort B (5 Capsules o.d.): PBO | Cohort C (4 Capsules b.i.d.): TIP | Cohort C (4 Capsules b.i.d.): TIP/PBO | Cohort C (4 Capsules b.i.d.): PBO | Total
Number analyzed (Participants) | 14 | 13 | 7 | 15 | 14 | 7 | 15 | 15 | 7 | 107
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.4 (12.66) | 57.5 (11.83) | 61.3 (7.45) | 64.3 (17.86) | 62.4 (16.71) | 69.1 (13.21) | 66.1 (12.23) | 60.8 (12.94) | 71.3 (10.39) | 63.4 (13.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 3 | 10 | 7 | 6 | 9 | 8 | 4 | 66
  Male | 5 | 3 | 4 | 5 | 7 | 1 | 6 | 7 | 3 | 41
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 12 | 11 | 7 | 13 | 11 | 5 | 15 | 15 | 7 | 96
  Asian | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
  Pacific Islander | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Other | 1 | 2 | 0 | 1 | 3 | 1 | 0 | 0 | 0 | 8

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Day 29 in Pseudomonas Aeruginosa (P. Aeruginosa) Density in Sputum (log10 CFUs)
Description: Microbiological data was collected to understand the direct impact of the drug on the pathogens. Sputum samples were cultured for the presence of three Pseudomonas aeruginosa (P. aeruginosa) biotypes measured were mucoid, dry and small colony variant. Change was determined using the formula = (Post-baseline value - baseline value). If no P. aeruginosa was isolated for a visit, log10 colony forming units (CFU) was imputed with log10 (19) for all biotypes. Only values for all morphotypes presented.
Time Frame: Baseline (Visit 101/Day 1), Visit 102 (Day 8), Visit 103 (Day 29)
Population: Full Analysis Set. Only the participants who had microbiological data at specified time points were included.
Measure: Mean (Standard Deviation); unit: log10 CFUs
Groups:
- Pooled TIP: Pooled Tobramycin inhalation powder (TIP): For efficacy analysis, subjects assigned to TIP groups were pooled across the 3 cohorts.
- Pooled TIP/PBO: Pooled Tobramycin inhalation powder (TIP) and inhaled placebo (PBO) cyclical: For efficacy analysis, subjects assigned to TIP/PBO groups were pooled across the 3 cohorts.
- Pooled PBO: Pooled inhaled placebo (PBO): For efficacy analysis, subjects assigned to Placebo groups were pooled across the 3 cohorts, as the number of placebo capsules was not expected to impact the efficacy assessments.
Arm/Group | Cohort A (3 Capsules o.d.): TIP | Cohort A (3 Capsules o.d.): TIP/PBO | Cohort B (5 Capsules o.d.): TIP | Cohort B (5 Capsules o.d.): TIP/PBO | Cohort C (4 Capsules b.i.d.): TIP | Cohort C (4 Capsules b.i.d.): TIP/PBO | Pooled TIP | Pooled TIP/PBO | Pooled PBO
Number analyzed (Participants) | 14 | 13 | 15 | 14 | 15 | 15 | 44 | 42 | 21
log10 CFUs
  Baseline: number analyzed (Participants) | 14 | 13 | 14 | 13 | 15 | 15 | 43 | 41 | 21
  Baseline | 6.80 (1.202) | 7.67 (1.507) | 6.10 (2.419) | 6.98 (1.804) | 6.79 (0.908) | 5.73 (1.885) | 6.57 (1.625) | 6.74 (1.892) | 7.09 (2.012)
  Change from BL at Day 8: number analyzed (Participants) | 10 | 11 | 9 | 12 | 13 | 10 | 32 | 33 | 21
  Change from BL at Day 8 | -2.82 (1.440) | -3.23 (2.204) | -2.04 (2.274) | -3.98 (1.865) | -4.54 (1.283) | -3.47 (1.583) | -3.30 (1.937) | -3.58 (1.878) | -0.72 (1.765)
  Change from BL at Day 29: number analyzed (Participants) | 14 | 10 | 9 | 10 | 13 | 12 | 36 | 32 | 21
  Change from BL at Day 29 | -2.61 (2.600) | -2.80 (2.823) | -1.56 (2.885) | -3.57 (2.218) | -4.36 (1.101) | -2.58 (2.871) | -2.98 (2.474) | -2.96 (2.618) | 0.05 (1.518)
Statistical Analysis 1: Comparison: Cohort A (3 Capsules o.d.): TIP vs Pooled PBO; Day 8 Cohort A: TIP, Pooled PBO; Test type: Other; LS Mean Diff (SE) vs pooled placebo = -2.4, 95% CI 2-sided [-3.62 to -1.22], Standard Error of Mean 0.60
Statistical Analysis 2: Comparison: Cohort A (3 Capsules o.d.): TIP/PBO vs Pooled PBO; Day 8 Cohort A: TIP/PBO, Pooled PBO; Test type: Other; LS Mean Diff (SE) vs pooled placebo = -2.1, 95% CI 2-sided [-3.30 to -0.98], Standard Error of Mean 0.58
Statistical Analysis 3: Comparison: Cohort B (5 Capsules o.d.): TIP vs Pooled PBO; Day 8 Cohort B: TIP, Pooled PBO; Test type: Other; LS Mean Diff (SE) vs pooled placebo = -1.9, 95% CI 2-sided [-3.20 to -0.68], Standard Error of Mean 0.63
Statistical Analysis 4: Comparison: Cohort B (5 Capsules o.d.): TIP/PBO vs Pooled PBO; Day 8 Cohort B: TIP/PBO, Pooled PBO; Test type: Other; LS Mean Diff (SE) vs pooled placebo = -3.3, 95% CI 2-sided [-4.38 to -2.15], Standard Error of Mean 0.56; LS Mean Diff (SE) vs pooled placebo
Statistical Analysis 5: Comparison: Cohort C (4 Capsules b.i.d.): TIP vs Pooled PBO; Day 8 Cohort C: TIP, Pooled PBO; Test type: Other; LS Mean Diff (SE) vs pooled placebo = -4.0, 95% CI 2-sided [-5.06 to -2.88], Standard Error of Mean 0.55
Statistical Analysis 6: Comparison: Cohort C (4 Capsules b.i.d.): TIP/PBO vs Pooled PBO; Day 8 Cohort C: TIP/PBO, Pooled PBO; Test type: Other; LS Mean Diff (SE) vs pooled placebo = -3.4, 95% CI 2-sided [-4.57 to -2.14], Standard Error of Mean 0.61
Statistical Analysis 7: Comparison: Pooled TIP vs Pooled PBO; Day 8: Pooled TIP, Pooled PBO; Test type: Other; LS Mean Diff (SE) vs pooled placebo = -2.8, 95% CI 2-sided [-3.66 to -1.89], Standard Error of Mean 0.44
Statistical Analysis 8: Comparison: Pooled TIP/PBO vs Pooled PBO; Day 8: Pooled TIP/PBO, Pooled PBO; Test type: Other; LS Mean Diff (SE) vs pooled placebo = -2.9, 95% CI 2-sided [-3.79 to -2.05], Standard Error of Mean 0.43
Statistical Analysis 9: Comparison: Cohort A (3 Capsules o.d.): TIP vs Pooled PBO; Day 29 Cohort A: TIP, Pooled PBO; Test type: Other; LS Mean Diff (SE) vs pooled placebo = -2.8, 95% CI 2-sided [-4.28 to -1.31], Standard Error of Mean 0.75
Statistical Analysis 10: Comparison: Cohort A (3 Capsules o.d.): TIP/PBO vs Pooled PBO; Day 29 Cohort A: TIP/PBO, Pooled PBO; Test type: Other; LS Mean Diff (SE) vs pooled placebo = -2.4, 95% CI 2-sided [-4.03 to -0.67], Standard Error of Mean 0.84
Statistical Analysis 11: Comparison: Cohort B (5 Capsules o.d.): TIP vs Pooled PBO; Day 29 Cohort B: TIP, Pooled PBO; Test type: Other; LS Mean Diff (SE) vs pooled placebo = -2.3, 95% CI 2-sided [-4.04 to -0.52], Standard Error of Mean 0.88
Statistical Analysis 12: Comparison: Cohort B (5 Capsules o.d.): TIP/PBO vs Pooled PBO; Day 29 Cohort B: TIP/PBO, Pooled PBO; Test type: Other; LS Mean Diff (SE) vs pooled placebo = -3.5, 95% CI 2-sided [-5.16 to -1.85], Standard Error of Mean 0.83
Statistical Analysis 13: Comparison: Cohort C (4 Capsules b.i.d.): TIP vs Pooled PBO; Day 29 Cohort C: TIP, Pooled PBO; Test type: Other; LS Mean Diff (SE) vs pooled placebo = -4.6, 95% CI 2-sided [-6.13 to -3.09], Standard Error of Mean 0.76
Statistical Analysis 14: Comparison: Cohort C (4 Capsules b.i.d.): TIP/PBO vs Pooled PBO; Day 29 Cohort C: TIP/PBO, Pooled PBO; Test type: Other; LS Mean Diff (SE) vs pooled placebo = -3.1, 95% CI 2-sided [-4.68 to -1.52], Standard Error of Mean 0.79
Statistical Analysis 15: Comparison: Pooled TIP vs Pooled PBO; Day 29: Pooled TIP, Pooled PBO; Test type: Other; LS Mean Diff (SE) vs pooled placebo = -3.2, 95% CI 2-sided [-4.43 to -2.02], Standard Error of Mean 0.61
Statistical Analysis 16: Comparison: Pooled TIP/PBO vs Pooled PBO; Day 29: Pooled TIP/PBO, Pooled PBO; Test type: Other; LS Mean Diff (SE) vs pooled placebo = -3.0, 95% CI 2-sided [-4.19 to -1.78], Standard Error of Mean 0.61

2. Secondary Outcome: Change From Baseline to Each Post-baseline Visit in Pseudomonas Aeruginosa (P. Aeruginosa) Density in Sputum (log10 CFUs)
Description: Microbiological data was collected to understand the direct impact of the drug on the pathogens. Sputum samples were cultured for the presence of three Pseudomonas aeruginosa (P. aeruginosa) biotypes measured were mucoid, dry and small colony variant. Change was determined using the formula = (Post-baseline value - baseline value). If no P. aeruginosa was isolated for a visit, log10 colony forming units (CFU) was imputed with log10 (19) for all biotypes. Only values for all morphotypes are presented.
Time Frame: Baseline (Visit 101/Day 1), Visit 104 (Day 57), Visit 105 (Day 85), Visit 106 (Day 113), End of Treatment (EOT), Visit 201 (Day 141), Visit 202 (Day 169)
Population: Full Analysis Set. Only the participants who had microbiological data at specified time points were included.
Measure: Mean (Standard Deviation); unit: log10 CFUs
Arm/Group | Cohort A (3 Capsules o.d.): TIP | Cohort A (3 Capsules o.d.): TIP/PBO | Cohort B (5 Capsules o.d.): TIP | Cohort B (5 Capsules o.d.): TIP/PBO | Cohort C (4 Capsules b.i.d.): TIP | Cohort C (4 Capsules b.i.d.): TIP/PBO | Pooled TIP | Pooled TIP/PBO | Pooled PBO
Number analyzed (Participants) | 14 | 13 | 15 | 14 | 15 | 15 | 44 | 42 | 21
log10 CFUs
  Baseline (BL): number analyzed (Participants) | 14 | 13 | 14 | 13 | 15 | 15 | 43 | 41 | 21
  Baseline (BL) | 6.80 (1.202) | 7.67 (1.507) | 6.10 (2.419) | 6.98 (1.804) | 6.79 (0.908) | 5.73 (1.885) | 6.57 (1.625) | 6.74 (1.892) | 7.09 (2.012)
  Change from BL at Day 57: number analyzed (Participants) | 11 | 11 | 8 | 11 | 13 | 10 | 32 | 32 | 17
  Change from BL at Day 57 | -1.72 (3.066) | -0.72 (2.677) | -0.90 (1.894) | -1.62 (2.804) | -3.53 (2.220) | -0.49 (2.305) | -2.25 (2.646) | -0.96 (2.576) | 0.20 (1.408)
  Change from BL at Day 85: number analyzed (Participants) | 11 | 9 | 6 | 10 | 9 | 8 | 26 | 27 | 17
  Change from BL at Day 85 | -2.47 (2.446) | -2.94 (2.492) | -2.81 (3.653) | -3.88 (2.470) | -3.08 (1.624) | -2.00 (2.951) | -2.76 (2.446) | -3.01 (2.641) | -0.36 (2.238)
  Change from BL at Day 113: number analyzed (Participants) | 8 | 10 | 4 | 9 | 7 | 6 | 19 | 25 | 16
  Change from BL at Day 113 | -2.94 (1.977) | -1.03 (2.002) | -1.82 (2.331) | -1.99 (3.020) | -3.17 (2.378) | -1.54 (3.534) | -2.79 (2.141) | -1.50 (2.707) | -0.20 (1.513)
  Change from BL at EOT: number analyzed (Participants) | 12 | 11 | 11 | 12 | 12 | 13 | 35 | 36 | 21
  Change from BL at EOT | -2.49 (1.896) | -1.08 (1.907) | -0.84 (1.766) | -1.86 (2.607) | -2.60 (2.531) | -1.29 (3.300) | -2.01 (2.192) | -1.42 (2.650) | -0.34 (1.445)
  Change from BL at Day 141: number analyzed (Participants) | 11 | 11 | 6 | 11 | 9 | 7 | 26 | 29 | 17
  Change from BL at Day 141 | -0.90 (2.113) | -0.82 (2.117) | 0.10 (1.551) | -2.17 (2.863) | -0.92 (2.385) | -0.87 (3.640) | -0.68 (2.067) | -1.34 (2.793) | -0.06 (2.191)
  Change from BL at Day 169: number analyzed (Participants) | 10 | 10 | 7 | 8 | 6 | 7 | 23 | 25 | 18
  Change from BL at Day 169 | -0.62 (2.324) | -1.19 (1.885) | 0.46 (1.651) | -1.27 (2.684) | 0.62 (1.038) | 1.33 (4.219) | 0.03 (1.882) | -0.51 (3.036) | 0.62 (2.694)
Statistical Analysis 1: Comparison: Cohort A (3 Capsules o.d.): TIP vs Pooled PBO; Day 57 Cohort A: TIP, Pooled PBO; Test type: Other; LS Mean Diff (SE) vs pooled placebo = -2.1, 95% CI 2-sided [-3.82 to -0.36], Standard Error of Mean 0.87
Statistical Analysis 2: Comparison: Cohort A (3 Capsules o.d.): TIP/PBO vs Pooled PBO; Day 57 Cohort A: TIP/PBO, Pooled PBO; Test type: Other; LS Mean Diff (SE) vs pooled placebo = -0.5, 95% CI 2-sided [-2.21 to 1.29], Standard Error of Mean 0.88
Statistical Analysis 3: Comparison: Cohort B (5 Capsules o.d.): TIP vs Pooled PBO; Day 57 Cohort B: TIP, Pooled PBO; Test type: Other; LS Mean Diff (SE) vs pooled placebo = -1.9, 95% CI 2-sided [-3.87 to 0.08], Standard Error of Mean 0.99
Statistical Analysis 4: Comparison: Cohort B (5 Capsules o.d.): TIP/PBO vs Pooled PBO; Day 57 Cohort B: TIP/PBO, Pooled PBO; Test type: Other; LS Mean Diff (SE) vs pooled placebo = -1.6, 95% CI 2-sided [-3.34 to 0.16], Standard Error of Mean 0.88
Statistical Analysis 5: Comparison: Cohort C (4 Capsules b.i.d.): TIP vs Pooled PBO; Day 57 Cohort C: TIP, Pooled PBO; Test type: Other; LS Mean Diff (SE) vs pooled placebo = -3.9, 95% CI 2-sided [-5.50 to -2.22], Standard Error of Mean 0.82
Statistical Analysis 6: Comparison: Cohort C (4 Capsules b.i.d.): TIP/PBO vs Pooled PBO; Day 57 Cohort C: TIP/PBO, Pooled PBO; Test type: Other; LS Mean Diff (SE) vs pooled placebo = -1.4, 95% CI 2-sided [-3.26 to 0.41], Standard Error of Mean 0.92
Statistical Analysis 7: Comparison: Pooled TIP vs Pooled PBO; Day 57: Pooled TIP, Pooled PBO; Test type: Other; LS Mean Diff (SE) vs pooled placebo = -2.6, 95% CI 2-sided [-3.98 to -1.25], Standard Error of Mean 0.68
Statistical Analysis 8: Comparison: Pooled TIP/PBO vs Pooled PBO; Day 57: Pooled TIP/PBO, Pooled PBO; Test type: Other; LS Mean Diff (SE) vs pooled placebo = -1.2, 95% CI 2-sided [-2.50 to 0.19], Standard Error of Mean 0.67
Statistical Analysis 9: Comparison: Cohort A (3 Capsules o.d.): TIP vs Pooled PBO; Day 85 Cohort A: TIP, Pooled PBO; Test type: Other; LS Mean Diff (SE) vs pooled placebo = -2.2, 95% CI 2-sided [-4.00 to -0.38], Standard Error of Mean 0.90
Statistical Analysis 10: Comparison: Cohort A (3 Capsules o.d.): TIP/PBO vs Pooled PBO; Day 85 Cohort A: TIP/PBO, Pooled PBO; Test type: Other; LS Mean Diff (SE) vs pooled placebo = -1.8, 95% CI 2-sided [-3.81 to 0.13], Standard Error of Mean 0.99
Statistical Analysis 11: Comparison: Cohort B (5 Capsules o.d.): TIP vs Pooled PBO; Day 85 Cohort B: TIP, Pooled PBO; Test type: Other; LS Mean Diff (SE) vs pooled placebo = -2.7, 95% CI 2-sided [-4.96 to -0.53], Standard Error of Mean 1.11
Statistical Analysis 12: Comparison: Cohort B (5 Capsules o.d.): TIP/PBO vs Pooled PBO; Day 85 Cohort B: TIP/PBO, Pooled PBO; Test type: Other; LS Mean Diff (SE) vs pooled placebo = -3.6, 95% CI 2-sided [-5.44 to -1.73], Standard Error of Mean 0.93
Statistical Analysis 13: Comparison: Cohort C (4 Capsules b.i.d.): TIP vs Pooled PBO; Day 85 Cohort C: TIP, Pooled PBO; Test type: Other; LS Mean Diff (SE) vs pooled placebo = -3.0, 95% CI 2-sided [-4.90 to -1.07], Standard Error of Mean 0.96
Statistical Analysis 14: Comparison: Cohort C (4 Capsules b.i.d.): TIP/PBO vs Pooled PBO; Day 85 Cohort C: TIP/PBO, Pooled PBO; Test type: Other; LS Mean Diff (SE) vs pooled placebo = -2.6, 95% CI 2-sided [-4.66 to -0.53], Standard Error of Mean 1.03
Statistical Analysis 15: Comparison: Pooled TIP vs Pooled PBO; Day 85: Pooled TIP, Pooled PBO; Test type: Other; LS Mean Diff (SE) vs pooled placebo = -2.6, 95% CI 2-sided [-4.11 to -1.17], Standard Error of Mean 0.74
Statistical Analysis 16: Comparison: Pooled TIP/PBO vs Pooled PBO; Day 85: Pooled TIP/PBO, Pooled PBO; Test type: Other; LS Mean Diff (SE) vs pooled placebo = -2.7, 95% CI 2-sided [-4.12 to -1.23], Standard Error of Mean 0.72
Statistical Analysis 17: Comparison: Cohort A (3 Capsules o.d.): TIP vs Pooled PBO; Day 113 Cohort A: TIP, Pooled PBO; Test type: Other; LS Mean Diff (SE) vs pooled placebo = -2.8, 95% CI 2-sided [-4.55 to -1.08], Standard Error of Mean 0.87
Statistical Analysis 18: Comparison: Cohort A (3 Capsules o.d.): TIP/PBO vs Pooled PBO; Day 113 Cohort A: TIP/PBO, Pooled PBO; Test type: Other; LS Mean Diff (SE) vs pooled placebo = 0.1, 95% CI 2-sided [-1.61 to 1.71], Standard Error of Mean 0.83
Statistical Analysis 19: Comparison: Cohort B (5 Capsules o.d.): TIP vs Pooled PBO; Day 113 Cohort B: TIP, Pooled PBO; Test type: Other; LS Mean Diff (SE) vs pooled placebo = -2.6, 95% CI 2-sided [-4.93 to -0.29], Standard Error of Mean 1.16
Statistical Analysis 20: Comparison: Cohort B (5 Capsules o.d.): TIP/PBO vs Pooled PBO; Day 113 Cohort B: TIP/PBO, Pooled PBO; Test type: Other; LS Mean Diff (SE) vs pooled placebo = -1.9, 95% CI 2-sided [-3.62 to -0.25], Standard Error of Mean 0.84
Statistical Analysis 21: Comparison: Cohort C (4 Capsules b.i.d.): TIP vs Pooled PBO; Day 113 Cohort C: TIP, Pooled PBO; Test type: Other; LS Mean Diff (SE) vs pooled placebo = -3.1, 95% CI 2-sided [-4.94 to -1.30], Standard Error of Mean 0.91
Statistical Analysis 22: Comparison: Cohort C (4 Capsules b.i.d.): TIP/PBO vs Pooled PBO; Day 113 Cohort C: TIP/PBO, Pooled PBO; Test type: Other; LS Mean Diff (SE) vs pooled placebo = -2.4, 95% CI 2-sided [-4.37 to -0.43], Standard Error of Mean 0.98
Statistical Analysis 23: Comparison: Pooled TIP vs Pooled PBO; Day 113: Pooled TIP, Pooled PBO; Test type: Other; LS Mean Diff (SE) vs pooled placebo = -2.8, 95% CI 2-sided [-4.24 to -1.45], Standard Error of Mean 0.70
Statistical Analysis 24: Comparison: Pooled TIP/PBO vs Pooled PBO; Day 113: Pooled TIP/PBO, Pooled PBO; Test type: Other; LS Mean Diff (SE) vs pooled placebo = -1.4, 95% CI 2-sided [-2.73 to -0.13], Standard Error of Mean 0.65
Statistical Analysis 25: Comparison: Cohort A (3 Capsules o.d.): TIP vs Pooled PBO; EoT Cohort A: TIP, Pooled PBO; Test type: Other; LS Mean Diff (SE) vs pooled placebo = -2.2, 95% CI 2-sided [-3.64 to -0.73], Standard Error of Mean 0.73
Statistical Analysis 26: Comparison: Cohort A (3 Capsules o.d.): TIP/PBO vs Pooled PBO; EoT Cohort A: TIP/PBO, Pooled PBO; Test type: Other; LS Mean Diff (SE) vs pooled placebo = -0.1, 95% CI 2-sided [-1.61 to 1.43], Standard Error of Mean 0.76
Statistical Analysis 27: Comparison: Cohort B (5 Capsules o.d.): TIP vs Pooled PBO; EoT Cohort B: TIP, Pooled PBO; Test type: Other; LS Mean Diff (SE) vs pooled placebo = -1.3, 95% CI 2-sided [-2.81 to 0.25], Standard Error of Mean 0.77
Statistical Analysis 28: Comparison: Cohort B (5 Capsules o.d.): TIP/PBO vs Pooled PBO; EoT Cohort B: TIP/PBO, Pooled PBO; Test type: Other; LS Mean Diff (SE) vs pooled placebo = -1.7, 95% CI 2-sided [-3.14 to -0.22], Standard Error of Mean 0.73
Statistical Analysis 29: Comparison: Cohort C (4 Capsules b.i.d.): TIP vs Pooled PBO; EoT Cohort C: TIP, Pooled PBO; Test type: Other; LS Mean Diff (SE) vs pooled placebo = -2.4, 95% CI 2-sided [-3.89 to -0.98], Standard Error of Mean 0.73
Statistical Analysis 30: Comparison: Cohort C (4 Capsules b.i.d.): TIP/PBO vs Pooled PBO; EoT Cohort C: TIP/PBO, Pooled PBO; Test type: Other; LS Mean Diff (SE) vs pooled placebo = -1.7, 95% CI 2-sided [-3.12 to -0.22], Standard Error of Mean 0.73
Statistical Analysis 31: Comparison: Pooled TIP vs Pooled PBO; EoT: Pooled TIP, Pooled PBO; Test type: Other; LS Mean Diff (SE) vs pooled placebo = -2.0, 95% CI 2-sided [-3.08 to -0.85], Standard Error of Mean 0.56
Statistical Analysis 32: Comparison: Pooled TIP/PBO vs Pooled PBO; EoT: Pooled TIP/PBO, Pooled PBO; Test type: Other; LS Mean Diff (SE) vs pooled placebo = -1.1, 95% CI 2-sided [-2.25 to -0.04], Standard Error of Mean 0.56
Statistical Analysis 33: Comparison: Cohort A (3 Capsules o.d.): TIP vs Pooled PBO; Day 141 Cohort A: TIP, Pooled PBO; Test type: Other; LS Mean Diff (SE) vs pooled placebo = -0.8, 95% CI 2-sided [-2.63 to 0.99], Standard Error of Mean 0.91
Statistical Analysis 34: Comparison: Cohort A (3 Capsules o.d.): TIP/PBO vs Pooled PBO; Day 141 Cohort A: TIP/PBO, Pooled PBO; Test type: Other; LS Mean Diff (SE) vs pooled placebo = 0.1, 95% CI 2-sided [-1.83 to 1.98], Standard Error of Mean 0.95
Statistical Analysis 35: Comparison: Cohort B (5 Capsules o.d.): TIP vs Pooled PBO; Day 141 Cohort B: TIP, Pooled PBO; Test type: Other; LS Mean Diff (SE) vs pooled placebo = 0.2, 95% CI 2-sided [-2.03 to 2.41], Standard Error of Mean 1.11
Statistical Analysis 36: Comparison: Cohort B (5 Capsules o.d.): TIP/PBO vs Pooled PBO; Day 141 Cohort B: TIP/PBO, Pooled PBO; Test type: Other; LS Mean Diff (SE) vs pooled placebo = -1.8, 95% CI 2-sided [-3.68 to -0.01], Standard Error of Mean 0.92
Statistical Analysis 37: Comparison: Cohort C (4 Capsules b.i.d.): TIP vs Pooled PBO; Day 141 Cohort C (4 capsules b.i.d.): TIP, Pooled PBO; Test type: Other; LS Mean Diff (SE) vs pooled placebo = -0.9, 95% CI 2-sided [-2.78 to 1.07], Standard Error of Mean 0.96
Statistical Analysis 38: Comparison: Cohort C (4 Capsules b.i.d.): TIP/PBO vs Pooled PBO; Day 141 Cohort C: TIP/PBO, Pooled PBO; Test type: Other; LS Mean Diff (SE) vs pooled placebo = -1.2, 95% CI 2-sided [-3.36 to 0.89], Standard Error of Mean 1.06
Statistical Analysis 39: Comparison: Pooled TIP vs Pooled PBO; Day 141: Pooled TIP, Pooled PBO; Test type: Other; LS Mean Diff (SE) vs pooled placebo = -0.5, 95% CI 2-sided [-1.97 to 0.98], Standard Error of Mean 0.74
Statistical Analysis 40: Comparison: Pooled TIP/PBO vs Pooled PBO; Day 141: Pooled TIP/PBO, Pooled PBO; Test type: Other; LS Mean Diff (SE) vs pooled placebo = -1.0, 95% CI 2-sided [-2.45 to 0.45], Standard Error of Mean 0.73
Statistical Analysis 41: Comparison: Cohort A (3 Capsules o.d.): TIP vs Pooled PBO; Day 169 Cohort A: TIP, Pooled PBO; Test type: Other; LS Mean Diff (SE) vs pooled placebo = -1.3, 95% CI 2-sided [-3.24 to 0.61], Standard Error of Mean 0.96
Statistical Analysis 42: Comparison: Cohort A (3 Capsules o.d.): TIP/PBO vs Pooled PBO; Day 169 Cohort A: TIP/PBO, Pooled PBO; Test type: Other; LS Mean Diff (SE) vs pooled placebo = -1.1, 95% CI 2-sided [-3.05 to 0.91], Standard Error of Mean 0.99
Statistical Analysis 43: Comparison: Cohort B (5 Capsules o.d.): TIP vs Pooled PBO; Day 169 Cohort B: TIP, Pooled PBO; Test type: Other; LS Mean Diff (SE) vs pooled placebo = -0.6, 95% CI 2-sided [-2.73 to 1.62], Standard Error of Mean 1.09
Statistical Analysis 44: Comparison: Cohort B (5 Capsules o.d.): TIP/PBO vs Pooled PBO; Day 169 Cohort B: TIP/PBO, Pooled PBO; Test type: Other; LS Mean Diff (SE) vs pooled placebo = -2.1, 95% CI 2-sided [-4.22 to -0.08], Standard Error of Mean 1.03
Statistical Analysis 45: Comparison: Cohort C (4 Capsules b.i.d.): TIP vs Pooled PBO; Day 169 Cohort C: TIP, Pooled PBO; Test type: Other; LS Mean Diff (SE) vs pooled placebo = -0.2, 95% CI 2-sided [-2.48 to 2.10], Standard Error of Mean 1.14
Statistical Analysis 46: Comparison: Cohort C (4 Capsules b.i.d.): TIP/PBO vs Pooled PBO; Day 169 Cohort C: TIP/PBO, Pooled PBO; Test type: Other; LS Mean Diff (SE) vs pooled placebo = -0.1, 95% CI 2-sided [-2.33 to 2.13], Standard Error of Mean 1.12
Statistical Analysis 47: Comparison: Pooled TIP vs Pooled PBO; Day 169: Pooled TIP, Pooled PBO; Test type: Other; LS Mean Diff (SE) vs pooled placebo = -0.7, 95% CI 2-sided [-2.24 to 0.86], Standard Error of Mean 0.77
Statistical Analysis 48: Comparison: Pooled TIP/PBO vs Pooled PBO; Day 169: Pooled TIP/PBO, Pooled PBO; Test type: Other; LS Mean Diff (SE) vs pooled placebo = -1.1, 95% CI 2-sided [-2.61 to 0.40], Standard Error of Mean 0.75

3. Secondary Outcome: Time to First Onset of Pulmonary Exacerbation by Exacerbation Category
Description: The time to first onset of pulmonary exacerbation compared to placebo was analyzed. Participants with pulmonary exacerbation were categorized as: a) Overall, b) Category 1 (Oral): treated with oral antibiotics only and c) Category 2 (Parenteral): treated with parenteral Antibiotics and/or requiring hospitalization. Participants were censored at the time of completion of study or early discontinuation if they did not have a pulmonary exacerbation during the study period.
Time Frame: Baseline (Visit 101/Day 1) to Visit 202 (Day 169)
Population: Full Analysis Set
Measure: Median (Full Range); unit: Days
Arm/Group | Cohort A (3 Capsules o.d.): TIP | Cohort A (3 Capsules o.d.): TIP/PBO | Cohort B (5 Capsules o.d.): TIP | Cohort B (5 Capsules o.d.): TIP/PBO | Cohort C (4 Capsules b.i.d.): TIP | Cohort C (4 Capsules b.i.d.): TIP/PBO | Pooled TIP | Pooled TIP/PBO | Pooled PBO
Number analyzed (Participants) | 14 | 13 | 15 | 14 | 15 | 15 | 44 | 42 | 21
Days
  Overall: number analyzed (Participants) | 6 | 4 | 5 | 5 | 4 | 6 | 15 | 15 | 10
  Overall | NA [39.00 to NA] — NA: Not estimable due to insufficient number of participants with events | NA [48.00 to NA] — NA: Not estimable due to insufficient number of participants with events | NA [15.00 to NA] — NA: Not estimable due to insufficient number of participants with events | NA [85.00 to NA] — NA: Not estimable due to insufficient number of participants with events | NA [127.00 to NA] — NA: Not estimable due to insufficient number of participants with events | NA [24.00 to NA] — NA: Not estimable due to insufficient number of participants with events | NA [127.00 to NA] — NA: Not estimable due to insufficient number of participants with events | NA [85.00 to NA] — NA: Not estimable due to insufficient number of participants with events | 173.00 [77.00 to NA] — NA: Not estimable due to insufficient number of participants with events
  Oral: number analyzed (Participants) | 2 | 4 | 3 | 4 | 1 | 3 | 6 | 11 | 8
  Oral | NA [NA to NA] — NA: Not estimable due to insufficient number of participants with events | NA [48.00 to NA] — NA: Not estimable due to insufficient number of participants with events | NA [22.00 to NA] — NA: Not estimable due to insufficient number of participants with events | NA [85.00 to NA] — NA: Not estimable due to insufficient number of participants with events | NA [NA to NA] — NA: Not estimable due to insufficient number of participants with events | NA [84.00 to NA] — NA: Not estimable due to insufficient number of participants with events | NA [NA to NA] — NA: Not estimable due to insufficient number of participants with events | NA [NA to NA] — NA: Not estimable due to insufficient number of participants with events | 173.00 [106.00 to NA] — NA: Not estimable due to insufficient number of participants with events
  Parenteral: number analyzed (Participants) | 4 | 0 | 2 | 2 | 1 | 4 | 7 | 6 | 1
  Parenteral | NA [110.00 to NA] — NA: Not estimable due to insufficient number of participants with events |  | NA [60.00 to NA] — NA: Not estimable due to insufficient number of participants with events | NA [154.00 to NA] — NA: Not estimable due to insufficient number of participants with events | NA [NA to NA] — NA: Not estimable due to insufficient number of participants with events | NA [33.00 to NA] — NA: Not estimable due to insufficient number of participants with events | NA [NA to NA] — NA: Not estimable due to insufficient number of participants with events | NA [NA to NA] — NA: Not estimable due to insufficient number of participants with events | NA [NA to NA] — NA: Not estimable due to insufficient number of participants with events
Statistical Analysis 1: Comparison: Cohort A (3 Capsules o.d.): TIP vs Pooled PBO; Overall Cohort A: TIP, Pooled PBO; Test type: Other; Hazard Ratio (HR) = 1.14, 95% CI 2-sided [0.14 to 3.18] — Based on Cox proportional hazards model with treatment as fixed effect and number of pulmonary exacerbations in the 12 months prior to screening as a covariate, stratified by baseline macrolide use
Statistical Analysis 2: Comparison: Cohort A (3 Capsules o.d.): TIP/PBO vs Pooled PBO; Overall Cohort A: TIP/PBO, Pooled PBO; Test type: Other; Hazard Ratio (HR) = 0.57, 95% CI 2-sided [0.18 to 1.85] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Cohort B (5 Capsules o.d.): TIP vs Pooled PBO; Overall Cohort B: TIP, Pooled PBO; Test type: Other; Hazard Ratio (HR) = 1.26, 95% CI 2-sided [0.42 to 3.77] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 4: Comparison: Cohort B (5 Capsules o.d.): TIP/PBO vs Pooled PBO; Overall Cohort B: TIP/PBO, Pooled PBO; Test type: Other; Hazard Ratio (HR) = 0.61, 95% CI 2-sided [0.20 to 1.83] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 5: Comparison: Cohort C (4 Capsules b.i.d.): TIP vs Pooled PBO; Overall Cohort C: TIP, Pooled PBO; Test type: Other; Hazard Ratio (HR) = 0.67, 95% CI 2-sided [0.21 to 2.17] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 6: Comparison: Cohort C (4 Capsules b.i.d.): TIP/PBO vs Pooled PBO; Overall Cohort C: TIP/PBO, Pooled PBO; Test type: Other; Hazard Ratio (HR) = 1.27, 95% CI 2-sided [0.44 to 3.62] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 7: Comparison: Pooled TIP vs Pooled PBO; Overall Pooled TIP, Pooled PBO; Test type: Other; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.44 to 2.23] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 8: Comparison: Pooled TIP/PBO vs Pooled PBO; Overall Pooled TIP/PBO, Pooled PBO; Test type: Other; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.34 to 1.71] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 9: Comparison: Cohort A (3 Capsules o.d.): TIP vs Pooled PBO; Oral Cohort A: TIP, Pooled PBO; Test type: Other; Hazard Ratio (HR) = 0.39, 95% CI 2-sided [0.08 to 1.83] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 10: Comparison: Cohort A (3 Capsules o.d.): TIP/PBO vs Pooled PBO; Oral Cohort A: TIP/PBO, Pooled PBO; Test type: Other; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.25 to 2.89] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 11: Comparison: Cohort B (5 Capsules o.d.): TIP vs Pooled PBO; Oral Cohort B: TIP, Pooled PBO; Test type: Other; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.25 to 3.93] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 12: Comparison: Cohort B (5 Capsules o.d.): TIP/PBO vs Pooled PBO; Oral Cohort B: TIP/PBO, Pooled PBO; Test type: Other; Hazard Ratio (HR) = 0.67, 95% CI 2-sided [0.19 to 2.36] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 13: Comparison: Cohort C (4 Capsules b.i.d.): TIP vs Pooled PBO; Oral Cohort C: TIP, Pooled PBO; Test type: Other; Hazard Ratio (HR) = 0.19, 95% CI 2-sided [0.02 to 1.57] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 14: Comparison: Cohort C (4 Capsules b.i.d.): TIP/PBO vs Pooled PBO; Oral Cohort C: TIP/PBO, Pooled PBO; Test type: Other; Hazard Ratio (HR) = 0.62, 95% CI 2-sided [0.16 to 2.41] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 15: Comparison: Pooled TIP vs Pooled PBO; Oral Pooled TIP, Pooled PBO; Test type: Other; Hazard Ratio (HR) = 0.42, 95% CI 2-sided [0.13 to 1.31] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 16: Comparison: Pooled TIP/PBO vs Pooled PBO; Oral Pooled TIP/PBO, Pooled PBO; Test type: Other; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.28 to 1.80] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 17: Comparison: Cohort A (3 Capsules o.d.): TIP vs Pooled PBO; Parenteral Cohort A: TIP, Pooled PBO; Test type: Other; Hazard Ratio (HR) = 10.71, 95% CI 2-sided [1.10 to 104.19] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 18: Comparison: Cohort B (5 Capsules o.d.): TIP vs Pooled PBO; Parenteral Cohort B: TIP, Pooled PBO; Test type: Other; Hazard Ratio (HR) = 4.62, 95% CI 2-sided [0.41 to 52.29] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 19: Comparison: Cohort B (5 Capsules o.d.): TIP/PBO vs Pooled PBO; Parenteral Cohort B: TIP/PBO, Pooled PBO; Test type: Other; Hazard Ratio (HR) = 3.23, 95% CI 2-sided [0.28 to 37.06] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 20: Comparison: Cohort C (4 Capsules b.i.d.): TIP vs Pooled PBO; Parenteral Cohort C: TIP, Pooled PBO; Test type: Other; Hazard Ratio (HR) = 1.61, 95% CI 2-sided [0.10 to 25.94] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 21: Comparison: Cohort C (4 Capsules b.i.d.): TIP/PBO vs Pooled PBO; Parenteral Cohort C: TIP/PBO, Pooled PBO; Test type: Other; Hazard Ratio (HR) = 11.30, 95% CI 2-sided [1.09 to 117.34] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 22: Comparison: Pooled TIP vs Pooled PBO; Parenteral Pooled TIP, Pooled PBO; Test type: Other; Hazard Ratio (HR) = 4.30, 95% CI 2-sided [0.50 to 37.32] — [estimate comment as in outcome 3, analysis 1]

4. Secondary Outcome: Duration of Pulmonary Exacerbation by Exacerbation Category
Description: The duration of pulmonary exacerbation compared to placebo was analyzed. Participants with pulmonary exacerbation were categorized as: a) Overall, b) Category 1 (Oral): treated with oral antibiotics only and c) Category 2 (Parenteral): treated with parenteral Antibiotics and/or requiring hospitalization.
Time Frame: Baseline (Visit 101/Day 1) to Visit 202 (Day 169)
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Cohort A (3 Capsules o.d.): TIP | Cohort A (3 Capsules o.d.): TIP/PBO | Cohort B (5 Capsules o.d.): TIP | Cohort B (5 Capsules o.d.): TIP/PBO | Cohort C (4 Capsules b.i.d.): TIP | Cohort C (4 Capsules b.i.d.): TIP/PBO | Pooled TIP | Pooled TIP/PBO | Pooled PBO
Number analyzed (Participants) | 14 | 13 | 15 | 14 | 15 | 15 | 44 | 42 | 21
Days
  Overall: number analyzed (Participants) | 10 | 8 | 6 | 7 | 4 | 8 | 20 | 23 | 13
  Overall | 15.7 (6.22) | 18.0 (8.26) | 20.2 (6.37) | 10.3 (5.12) | 25.5 (27.09) | 14.8 (6.73) | 19.0 (12.64) | 15.2 (7.39) | 14.5 (5.61)
  Oral: number analyzed (Participants) | 2 | 7 | 4 | 5 | 1 | 3 | 7 | 15 | 11
  Oral | 19.5 (12.02) | 15.4 (4.24) | 19.3 (3.20) | 8.3 (4.16) | 14.0 (NA) — NA: Not estimable due to insufficient number of participants with events | 16.3 (5.51) | 18.6 (5.77) | 14.0 (5.24) | 15.6 (5.75)
  Parenteral: number analyzed (Participants) | 5 | 0 | 2 | 2 | 1 | 4 | 8 | 6 | 1
  Parenteral | 15.0 (5.52) |  | 22.0 (12.73) | 16.0 (NA) — NA: Not estimable due to insufficient number of participants with events | 66.0 (NA) — NA: Not estimable due to insufficient number of participants with events | 16.8 (4.86) | 23.1 (18.73) | 16.6 (4.22) | 10.0 (NA) — NA: Not estimable due to insufficient number of participants with events
Statistical Analysis 1: Comparison: Cohort A (3 Capsules o.d.): TIP vs Pooled PBO; Overall Cohort A: TIP, Pooled PBO; Test type: Other; LS Mean Diff (SE) vs pooled placebo = 9.8, 95% CI 2-sided [-27.15 to 46.81], Standard Error of Mean 18.15 — ANCOVA model includes treatment as a fixed-effect factor and number of pulmonary exacerbations in the 12 months prior to screening as a covariate
Statistical Analysis 2: Comparison: Cohort A (3 Capsules o.d.): TIP/PBO vs Pooled PBO; Overall Cohort A: TIP/PBO, Pooled PBO; Test type: Other; LS Mean Diff (SE) vs pooled placebo = 19.8, 95% CI 2-sided [-22.63 to 62.14], Standard Error of Mean 20.81 — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Cohort B (5 Capsules o.d.): TIP vs Pooled PBO; Overall Cohort B: TIP, Pooled PBO; Test type: Other; LS Mean Diff (SE) vs pooled placebo = 8.0, 95% CI 2-sided [-31.32 to 47.26], Standard Error of Mean 19.29 — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 4: Comparison: Cohort B (5 Capsules o.d.): TIP/PBO vs Pooled PBO; Overall Cohort B: TIP/PBO, Pooled PBO; Test type: Other; LS Mean Diff (SE) vs pooled placebo = 12.7, 95% CI 2-sided [-26.49 to 51.89], Standard Error of Mean 19.24 — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 5: Comparison: Cohort C (4 Capsules b.i.d.): TIP vs Pooled PBO; Overall Cohort C: TIP, Pooled PBO; Test type: Other; LS Mean Diff (SE) vs pooled placebo = 46.5, 95% CI 2-sided [3.37 to 89.61], Standard Error of Mean 21.17 — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 6: Comparison: Cohort C (4 Capsules b.i.d.): TIP/PBO vs Pooled PBO; Overall Cohort C: TIP/PBO, Pooled PBO; Test type: Other; LS Mean Diff (SE) vs pooled placebo = 3.2, 95% CI 2-sided [-34.21 to 40.64], Standard Error of Mean 18.37 — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 7: Comparison: Pooled TIP vs Pooled PBO; Overall Pooled TIP, Pooled PBO; Test type: Other; LS Mean Diff (SE) vs pooled placebo = 21.4, 95% CI 2-sided [-8.03 to 50.89], Standard Error of Mean 14.46 — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 8: Comparison: Pooled TIP/PBO vs Pooled PBO; Overall Pooled TIP/PBO, Pooled PBO; Test type: Other; LS Mean Diff (SE) vs pooled placebo = 11.9, 95% CI 2-sided [-17.52 to 41.29], Standard Error of Mean 14.44 — [estimate comment as in outcome 4, analysis 1]

5. Secondary Outcome: Exposure Adjusted Rate of Pulmonary Exacerbations (PE) Over the Entire Study Period
Description: The exposure adjusted rate of pulmonary exacerbation compared to placebo was analyzed. Participants with pulmonary exacerbation were categorized as: a) Overall, b) Category 1 (Oral): treated with oral antibiotics only and c) Category 2 (Parenteral): treated with parenteral Antibiotics and/or requiring hospitalization. The Exposure adjusted rate = (Number of pulmonary exacerbations reported during the study period) / (sum of study duration in days for all participants/ 365.25). Only descriptive analysis performed.
Time Frame: Baseline (Visit 101/Day 1) to Visit 202 (Day 169)
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: pulmonary exacerbation per study years
Arm/Group | Cohort A (3 Capsules o.d.): TIP | Cohort A (3 Capsules o.d.): TIP/PBO | Cohort B (5 Capsules o.d.): TIP | Cohort B (5 Capsules o.d.): TIP/PBO | Cohort C (4 Capsules b.i.d.): TIP | Cohort C (4 Capsules b.i.d.): TIP/PBO | Pooled TIP | Pooled TIP/PBO | Pooled PBO
Number analyzed (Participants) | 14 | 13 | 15 | 14 | 15 | 15 | 44 | 42 | 21
pulmonary exacerbation per study years
  Overall: number analyzed (Participants) | 6 | 4 | 5 | 5 | 4 | 6 | 15 | 15 | 10
  Overall | 1.71 [0.92 to 3.17] | 1.39 [0.70 to 2.78] | 1.29 [0.58 to 2.87] | 1.20 [0.57 to 2.51] | 0.66 [0.25 to 1.76] | 1.46 [0.73 to 2.93] | 1.21 [0.78 to 1.87] | 1.35 [0.90 to 2.03] | 1.41 [0.82 to 2.42]
  Oral: number analyzed (Participants) | 2 | 4 | 3 | 4 | 1 | 3 | 6 | 11 | 8
  Oral | 0.34 [0.09 to 1.37] | 1.22 [0.58 to 2.56] | 0.86 [0.32 to 2.29] | 0.85 [0.36 to 2.05] | 0.16 [0.02 to 1.17] | 0.55 [0.18 to 1.70] | 0.42 [0.20 to 0.89] | 0.88 [0.53 to 1.46] | 1.19 [0.66 to 2.15]
  Parenteral: number analyzed (Participants) | 4 | 0 | 2 | 2 | 1 | 4 | 7 | 6 | 1
  Parenteral | 0.85 [0.36 to 2.05] |  | 0.43 [0.11 to 1.72] | 0.34 [0.09 to 1.37] | 0.16 [0.02 to 1.17] | 0.73 [0.27 to 1.95] | 0.48 [0.24 to 0.96] | 0.35 [0.16 to 0.78] | 0.11 [0.02 to 0.77]

6. Secondary Outcome: Percentage of Participants With at Least One Pulmonary Exacerbation by Exacerbation Category
Description: Pulmonary exacerbations are defined as events requiring antibiotic therapy AND for which at least 3 of the following 6 symptoms, signs, or findings were present outside of normal variation: 1. Increased sputum volume, or change in viscosity/consistency or purulence for more than 24 hours; 2. Increased shortness of breath at rest or on exercise for more than 24 hours; 3. Increased cough for more than 24 hours; 4. Fever of ≥38° Celsius within the last 24 hours; 5. Increased malaise/fatigue/lethargy for more than 24 hours; 6. A reduction in forced expiratory volume in the first second of expiration (FEV1) or forced vital capacity (FVC) of least 10% from screening.
  Participants were categorized as: a) Overall, b) Category 1: treated with oral antibiotics only and c) Category 2: treated with parenteral Antibiotics and/or requiring hospitalization.
  Only descriptive analysis performed.
Time Frame: Baseline (Visit 101/Day 1) to Visit 202 (Day 169)
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A (3 Capsules o.d.): TIP | Cohort A (3 Capsules o.d.): TIP/PBO | Cohort B (5 Capsules o.d.): TIP | Cohort B (5 Capsules o.d.): TIP/PBO | Cohort C (4 Capsules b.i.d.): TIP | Cohort C (4 Capsules b.i.d.): TIP/PBO | Pooled TIP | Pooled TIP/PBO | Pooled PBO
Number analyzed (Participants) | 14 | 13 | 15 | 14 | 15 | 15 | 44 | 42 | 21
Participants
  Overall: No of participants with no events | 8 | 9 | 10 | 9 | 11 | 9 | 29 | 27 | 11
  Overall: No. of participants with 1 event | 3 | 1 | 4 | 3 | 4 | 4 | 11 | 8 | 7
  Overall: No. of participants with 2 events | 2 | 2 | 1 | 2 | 0 | 2 | 3 | 6 | 3
  Overall: No. of participants with 3 events | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0
  Oral: No of participants with no events | 12 | 9 | 12 | 10 | 14 | 12 | 38 | 31 | 13
  Oral: No. of participants with 1 event | 2 | 2 | 2 | 3 | 1 | 3 | 5 | 8 | 5
  Oral: No. of participants with 2 events | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 2 | 3
  Oral: No. of participants with 3 events | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Parenteral: No of participants with no events | 10 | 13 | 13 | 12 | 14 | 11 | 37 | 36 | 20
  Parenteral: No. of participants with 1 event | 3 | 0 | 2 | 2 | 1 | 4 | 6 | 6 | 1
  Parenteral: No. of participants with 2 events | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Parenteral: No. of participants with 3 events | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Percentage of Participants Who Permanently Discontinued Study Drug Due to Pulmonary Exacerbation
Description: The percentage of participants who permanently discontinued study drug due to pulmonary exacerbation compared to placebo was analyzed.
Time Frame: Baseline (Visit 101/Day 1) to Visit 202 (Day 169)
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A (3 Capsules o.d.): TIP | Cohort A (3 Capsules o.d.): TIP/PBO | Cohort B (5 Capsules o.d.): TIP | Cohort B (5 Capsules o.d.): TIP/PBO | Cohort C (4 Capsules b.i.d.): TIP | Cohort C (4 Capsules b.i.d.): TIP/PBO | Pooled TIP | Pooled TIP/PBO | Pooled PBO
Number analyzed (Participants) | 14 | 13 | 15 | 14 | 15 | 15 | 44 | 42 | 21
Participants | 2 | 0 | 1 | 0 | 0 | 2 | 41 | 40 | 0

8. Secondary Outcome: Time to Permanent Study Drug Discontinuation Due to Pulmonary Exacerbation
Description: The time to permanent study drug discontinuation due to Pulmonary exacerbation. Participants were censored at the time of last contact if they did not permanently discontinue study drug due to pulmonary exacerbation requiring during the study period. Only descriptive analysis performed.
Time Frame: Baseline (Visit 101/Day 1) to Visit 202 (Day 169)
Population: Full Analysis Set
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Cohort A (3 Capsules o.d.): TIP | Cohort A (3 Capsules o.d.): TIP/PBO | Cohort B (5 Capsules o.d.): TIP | Cohort B (5 Capsules o.d.): TIP/PBO | Cohort C (4 Capsules b.i.d.): TIP | Cohort C (4 Capsules b.i.d.): TIP/PBO | Pooled TIP | Pooled TIP/PBO | Pooled PBO
Number analyzed (Participants) | 14 | 13 | 15 | 14 | 15 | 15 | 44 | 42 | 21
Days | NA [94.00 to NA] — NA: Not estimable due to insufficient number of participants with events | NA [NA to NA] — NA: Not estimable due to insufficient number of participants with events | NA [NA to NA] — NA: Not estimable due to insufficient number of participants with events | NA [NA to NA] — NA: Not estimable due to insufficient number of participants with events | NA [NA to NA] — NA: Not estimable due to insufficient number of participants with events | NA [84.00 to NA] — NA: Not estimable due to insufficient number of participants with events | NA [NA to NA] — NA: Not estimable due to insufficient number of participants with events | NA [NA to NA] — NA: Not estimable due to insufficient number of participants with events | NA [NA to NA] — NA: Not estimable due to insufficient number of participants with events

9. Secondary Outcome: Time to First Use (Overall, Oral, and Parenteral) of Anti-pseudomonal Antibiotics Usage
Description: The time to first use of anti-pseudomonal antibiotics administered compared to placebo was analyzed. Participants were censored at the time of last contact if they did not have anti-pseudomonal antibiotics over the entire study period.
Time Frame: From Baseline (Visit 101/Day 1) up to approximately Day 173
Population: Full Analysis Set. Only the participants who required antipseudomonal antibiotics were included.
Measure: Median (Full Range); unit: Days
Arm/Group | Cohort A (3 Capsules o.d.): TIP | Cohort A (3 Capsules o.d.): TIP/PBO | Cohort B (5 Capsules o.d.): TIP | Cohort B (5 Capsules o.d.): TIP/PBO | Cohort C (4 Capsules b.i.d.): TIP | Cohort C (4 Capsules b.i.d.): TIP/PBO | Pooled TIP | Pooled TIP/PBO | Pooled PBO
Number analyzed (Participants) | 14 | 13 | 15 | 14 | 15 | 15 | 44 | 42 | 21
Days
  Overall: number analyzed (Participants) | 8 | 4 | 6 | 7 | 3 | 7 | 17 | 18 | 12
  Overall | 122.00 [29.00 to NA] — NA: Not estimable due to insufficient number of participants with events | NA [50.00 to NA] — NA: Not estimable due to insufficient number of participants with events | 116.00 [17.00 to NA] — NA: Not estimable due to insufficient number of participants with events | 161.00 [58.00 to NA] — NA: Not estimable due to insufficient number of participants with events | NA [127.00 to NA] — NA: Not estimable due to insufficient number of participants with events | NA [11.00 to NA] — NA: Not estimable due to insufficient number of participants with events | NA [110.00 to NA] — NA: Not estimable due to insufficient number of participants with events | NA [84.00 to NA] — NA: Not estimable due to insufficient number of participants with events | 141.00 [57.00 to NA] — NA: Not estimable due to insufficient number of participants with events
  Oral: number analyzed (Participants) | 5 | 4 | 5 | 6 | 2 | 6 | 12 | 16 | 10
  Oral | NA [43.00 to NA] — NA: Not estimable due to insufficient number of participants with events | NA [50.00 to NA] — NA: Not estimable due to insufficient number of participants with events | NA [17.00 to NA] — NA: Not estimable due to insufficient number of participants with events | NA [85.00 to NA] — NA: Not estimable due to insufficient number of participants with events | NA [NA to NA] — NA: Not estimable due to insufficient number of participants with events | NA [11.00 to NA] — NA: Not estimable due to insufficient number of participants with events | NA [NA to NA] — NA: Not estimable due to insufficient number of participants with events | NA [85.00 to NA] — NA: Not estimable due to insufficient number of participants with events | 173.00 [106.00 to NA] — NA: Not estimable due to insufficient number of participants with events
  Parenteral: number analyzed (Participants) | 5 | 0 | 2 | 4 | 1 | 4 | 8 | 8 | 3
  Parenteral | NA [105.0 to NA] — NA: Not estimable due to insufficient number of participants with events |  | NA [63.00 to NA] — NA: Not estimable due to insufficient number of participants with events | NA [95.00 to NA] — NA: Not estimable due to insufficient number of participants with events | NA [NA to NA] — NA: Not estimable due to insufficient number of participants with events | NA [37.00 to NA] — NA: Not estimable due to insufficient number of participants with events | NA [NA to NA] — NA: Not estimable due to insufficient number of participants with events | NA [NA to NA] — NA: Not estimable due to insufficient number of participants with events | NA [NA to NA] — NA: Not estimable due to insufficient number of participants with events
Statistical Analysis 1: Comparison: Cohort A (3 Capsules o.d.): TIP vs Pooled PBO; Overall Cohort A: TIP, Pooled PBO; Test type: Other; Hazard Ratio (HR) = 1.26, 95% CI 2-sided [0.51 to 3.13] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Cohort A (3 Capsules o.d.): TIP/PBO vs Pooled PBO; Overall Cohort A: TIP/PBO, Pooled PBO; Test type: Other; Hazard Ratio (HR) = 0.47, 95% CI 2-sided [0.15 to 1.46] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Cohort B (5 Capsules o.d.): TIP vs Pooled PBO; Overall Cohort B: TIP, Pooled PBO; Test type: Other; Hazard Ratio (HR) = 1.18, 95% CI 2-sided [0.44 to 3.21] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 4: Comparison: Cohort B (5 Capsules o.d.): TIP/PBO vs Pooled PBO; Overall Cohort B: TIP/PBO, Pooled PBO; Test type: Other; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.32 to 2.18] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 5: Comparison: Cohort C (4 Capsules b.i.d.): TIP vs Pooled PBO; Overall Cohort C: TIP, Pooled PBO; Test type: Other; Hazard Ratio (HR) = 0.35, 95% CI 2-sided [0.10 to 1.27] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 6: Comparison: Cohort C (4 Capsules b.i.d.): TIP/PBO vs Pooled PBO; Overall Cohort C: TIP/PBO, Pooled PBO; Test type: Other; Hazard Ratio (HR) = 1.13, 95% CI 2-sided [0.43 to 2.99] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 7: Comparison: Pooled TIP vs Pooled PBO; Overall Pooled TIP, Pooled PBO; Test type: Other; Hazard Ratio (HR) = 0.81, 95% CI 2-sided [0.37 to 1.76] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 8: Comparison: Pooled TIP/PBO vs Pooled PBO; Overall Pooled TIP/PBO, Pooled PBO; Test type: Other; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.36 to 1.61] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 9: Comparison: Cohort A (3 Capsules o.d.): TIP vs Pooled PBO; Oral Cohort A: TIP, Pooled PBO; Test type: Other; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.30 to 2.55] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 10: Comparison: Cohort A (3 Capsules o.d.): TIP/PBO vs Pooled PBO; Oral Cohort A: TIP/PBO, Pooled PBO; Test type: Other; Hazard Ratio (HR) = 0.63, 95% CI 2-sided [0.20 to 2.03] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 11: Comparison: Cohort B (5 Capsules o.d.): TIP vs Pooled PBO; Oral Cohort B: TIP, Pooled PBO; Test type: Other; Hazard Ratio (HR) = 1.20, 95% CI 2-sided [0.40 to 3.60] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 12: Comparison: Cohort B (5 Capsules o.d.): TIP/PBO vs Pooled PBO; Oral Cohort B: TIP/PBO, Pooled PBO; Test type: Other; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.31 to 2.55] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 13: Comparison: Cohort C (4 Capsules b.i.d.): TIP vs Pooled PBO; Oral Cohort C: TIP, Pooled PBO; Test type: Other; Hazard Ratio (HR) = 0.28, 95% CI 2-sided [0.06 to 1.27] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 14: Comparison: Cohort C (4 Capsules b.i.d.): TIP/PBO vs Pooled PBO; Oral Cohort C: TIP/PBO, Pooled PBO; Test type: Other; Hazard Ratio (HR) = 1.30, 95% CI 2-sided [0.45 to 3.73] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 15: Comparison: Pooled TIP vs Pooled PBO; Oral Pooled TIP, Pooled PBO; Test type: Other; Hazard Ratio (HR) = 0.66, 95% CI 2-sided [0.27 to 1.60] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 16: Comparison: Pooled TIP/PBO vs Pooled PBO; Oral Pooled TIP/PBO, Pooled PBO; Test type: Other; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.40 to 2.02] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 17: Comparison: Cohort A (3 Capsules o.d.): TIP vs Pooled PBO; Parenteral Cohort A: TIP, Pooled PBO; Test type: Other; Hazard Ratio (HR) = 3.72, 95% CI 2-sided [0.84 to 16.52] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 18: Comparison: Cohort B (5 Capsules o.d.): TIP vs Pooled PBO; Parenteral Cohort B: TIP, Pooled PBO; Test type: Other; Hazard Ratio (HR) = 1.34, 95% CI 2-sided [0.22 to 8.16] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 19: Comparison: Cohort B (5 Capsules o.d.): TIP/PBO vs Pooled PBO; Parenteral Cohort B: TIP/PBO, Pooled PBO; Test type: Other; Hazard Ratio (HR) = 2.15, 95% CI 2-sided [0.46 to 10.05] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 20: Comparison: Cohort C (4 Capsules b.i.d.): TIP vs Pooled PBO; Parenteral Cohort C: TIP, Pooled PBO; Test type: Other; Hazard Ratio (HR) = 0.50, 95% CI 2-sided [0.05 to 4.87] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 21: Comparison: Cohort C (4 Capsules b.i.d.): TIP/PBO vs Pooled PBO; Parenteral Cohort C: TIP/PBO, Pooled PBO; Test type: Other; Hazard Ratio (HR) = 2.56, 95% CI 2-sided [0.53 to 12.49] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 22: Comparison: Pooled TIP vs Pooled PBO; Paremteral Pooled TIP, Pooled PBO; Test type: Other; Hazard Ratio (HR) = 1.36, 95% CI 2-sided [0.33 to 5.68] — [estimate comment as in outcome 3, analysis 1]

10. Secondary Outcome: Percentage of Participants Requiring Anti-pseudomonal Antibiotics
Description: The percentage of participants requiring anti-pseudomonal antibiotics compared to placebo was analyzed. Only descriptive analysis performed.
Time Frame: Baseline (Visit 101/Day 1) to Visit 202 (Day 169)
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A (3 Capsules o.d.): TIP | Cohort A (3 Capsules o.d.): TIP/PBO | Cohort B (5 Capsules o.d.): TIP | Cohort B (5 Capsules o.d.): TIP/PBO | Cohort C (4 Capsules b.i.d.): TIP | Cohort C (4 Capsules b.i.d.): TIP/PBO | Pooled TIP | Pooled TIP/PBO | Pooled PBO
Number analyzed (Participants) | 14 | 13 | 15 | 14 | 15 | 15 | 44 | 42 | 21
Participants
  Overall: Any anti-pseudomonal antibiotic use?=Yes | 8 | 4 | 6 | 7 | 3 | 7 | 17 | 18 | 12
  Overall: Any anti-pseudomonal antibiotic use?=No | 6 | 9 | 9 | 7 | 12 | 8 | 27 | 24 | 9
  Oral: Any anti-pseudomonal antibiotic use?=Yes | 5 | 4 | 5 | 6 | 2 | 6 | 12 | 16 | 10
  Oral: Any anti-pseudomonal antibiotic use?=No | 9 | 9 | 10 | 8 | 13 | 9 | 32 | 26 | 11
  Parenteral: Any anti-pseudomonal antibiotic use?=Yes | 5 | 0 | 2 | 4 | 1 | 4 | 8 | 8 | 3
  Parenteral: Any anti-pseudomonal antibiotic use?=No | 9 | 13 | 13 | 10 | 14 | 11 | 36 | 34 | 18

11. Secondary Outcome: Duration of Anti-pseudomonal Antibiotics Usage
Description: The total number of days of new anti-pseudomonal antibiotic use compared to placebo was analyzed. Only descriptive analysis
Time Frame: Baseline (Visit 101/Day 1) to Visit 202 (Day 169)
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Cohort A (3 Capsules o.d.): TIP | Cohort A (3 Capsules o.d.): TIP/PBO | Cohort B (5 Capsules o.d.): TIP | Cohort B (5 Capsules o.d.): TIP/PBO | Cohort C (4 Capsules b.i.d.): TIP | Cohort C (4 Capsules b.i.d.): TIP/PBO | Pooled TIP | Pooled TIP/PBO | Pooled PBO
Number analyzed (Participants) | 14 | 13 | 15 | 14 | 15 | 15 | 44 | 42 | 21
Days
  Overall: number analyzed (Participants) | 8 | 4 | 6 | 7 | 3 | 7 | 17 | 18 | 12
  Overall | 18.4 (10.39) | 20.0 (12.03) | 19.2 (14.84) | 25.7 (13.21) | 15.3 (10.07) | 15.7 (10.90) | 18.1 (11.43) | 20.6 (12.24) | 14.6 (8.27)
  Oral: number analyzed (Participants) | 5 | 4 | 5 | 6 | 2 | 6 | 12 | 16 | 10
  Oral | 14.2 (7.79) | 19.8 (12.34) | 15.0 (7.42) | 14.0 (10.92) | 20.0 (8.49) | 10.8 (6.24) | 15.5 (7.29) | 14.3 (9.79) | 13.7 (7.41)
  Parenteral: number analyzed (Participants) | 5 | 0 | 2 | 4 | 1 | 4 | 8 | 8 | 3
  Parenteral | 15.0 (10.02) |  | 20.0 (14.14) | 23.8 (15.20) | 6.0 (NA) — NA: Not estimable due to insufficient number of participants with events | 11.3 (2.75) | 15.1 (10.23) | 17.5 (12.12) | 12.7 (7.64)

12. Secondary Outcome: Percentage of Participants Requiring Hospitalization Due to Serious Respiratory-related Adverse Events
Description: The percentage of participants requiring hospitalization due to serious respiratory-related adverse events (other than those regularly scheduled hospitalization that were planned prior to study start) was analyzed to define severity of pulmonary exacerbations compared to placebo. Only descriptive analysis performed.
Time Frame: Baseline (Visit 101/Day 1) to Visit 202 (Day 169)
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A (3 Capsules o.d.): TIP | Cohort A (3 Capsules o.d.): TIP/PBO | Cohort B (5 Capsules o.d.): TIP | Cohort B (5 Capsules o.d.): TIP/PBO | Cohort C (4 Capsules b.i.d.): TIP | Cohort C (4 Capsules b.i.d.): TIP/PBO | Pooled TIP | Pooled TIP/PBO | Pooled PBO
Number analyzed (Participants) | 14 | 13 | 15 | 14 | 15 | 15 | 44 | 42 | 21
Participants
  No of participants with 0 event | 10 | 13 | 13 | 12 | 14 | 11 | 37 | 36 | 19
  No. of participants with 1 event | 3 | 0 | 2 | 1 | 0 | 4 | 5 | 5 | 2
  No. of participants with 2 events | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
  No. of participants with > 2 events | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0

13. Secondary Outcome: Duration of Hospitalization Due to Serious Respiratory-related Adverse Events
Description: The duration of hospitalization due to serious respiratory-related adverse events (other than those regularly scheduled hospitalization that were planned prior to study start) was analyzed to define severity of pulmonary exacerbations compared to placebo. Only descriptive analysis performed.
Time Frame: Baseline (Visit 101/Day 1) to Visit 202 (Day 169)
Population: Full Analysis Set. Only the participants with at least one hospitalization are included in the analysis
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Cohort A (3 Capsules o.d.): TIP | Cohort A (3 Capsules o.d.): TIP/PBO | Cohort B (5 Capsules o.d.): TIP | Cohort B (5 Capsules o.d.): TIP/PBO | Cohort C (4 Capsules b.i.d.): TIP | Cohort C (4 Capsules b.i.d.): TIP/PBO | Pooled TIP | Pooled TIP/PBO | Pooled PBO
Number analyzed (Participants) | 4 | 0 | 2 | 2 | 1 | 4 | 7 | 6 | 2
Days | 15.2 (5.19) |  | 22.0 (12.73) | 12.2 (6.06) | 11.0 (NA) — NA: Not estimable due to insufficient number of participants with events | 19.0 (5.23) | 16.2 (7.05) | 15.2 (6.44) | 10.5 (0.71)

14. Secondary Outcome: Number of Hospitalization Due to Serious Respiratory-related Adverse Events
Description: The number of hospitalization due to serious respiratory-related AEs was analyzed to define severity of pulmonary exacerbations compared to placebo. Respiratory related adverse events were identified using the AEs captured under system organ class 'Respiratory, thoracic and mediastinal disorders' and 'Infections and infestations'.
Time Frame: Baseline (Visit 101/Day 1) to Visit 202 (Day 169)
Population: Full Analysis Set
Measure: Number; unit: Hospitalization
Arm/Group | Cohort A (3 Capsules o.d.): TIP | Cohort A (3 Capsules o.d.): TIP/PBO | Cohort B (5 Capsules o.d.): TIP | Cohort B (5 Capsules o.d.): TIP/PBO | Cohort C (4 Capsules b.i.d.): TIP | Cohort C (4 Capsules b.i.d.): TIP/PBO | Pooled TIP | Pooled TIP/PBO | Pooled PBO
Number analyzed (Participants) | 14 | 13 | 15 | 14 | 15 | 15 | 44 | 42 | 21
Hospitalization | 6 | 0 | 2 | 5 | 2 | 4 | 10 | 9 | 2
Statistical Analysis 1: Comparison: Cohort A (3 Capsules o.d.): TIP vs Pooled PBO; Cohort A (3 capsules o.d.): TIP, Pooled PBO; Test type: Other; Odds Ratio, log = 5.62, 95% CI 2-sided [0.83 to 38.18] — Generalized linear model assuming the negative binomial distribution including treatment and baseline macrolide use as class-effect factors. The log exposure to study in years is included as an offset variable in the model
Statistical Analysis 2: Comparison: Cohort B (5 Capsules o.d.): TIP vs Pooled PBO; Cohort B (5 capsules o.d.): TIP, Pooled PBO; Test type: Other; Odds Ratio, log = 2.00, 95% CI 2-sided [0.21 to 19.16] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 3: Comparison: Cohort B (5 Capsules o.d.): TIP/PBO vs Pooled PBO; Cohort B (5 capsules o.d.): TIP/PBO, Pooled PBO; Test type: Other; Odds Ratio, log = 3.05, 95% CI 2-sided [0.43 to 21.80] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 4: Comparison: Cohort C (4 Capsules b.i.d.): TIP vs Pooled PBO; Cohort C (4 capsules b.i.d.): TIP, Pooled PBO; Test type: Other; Odds Ratio, log = 1.84, 95% CI 2-sided [0.19 to 17.42] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 5: Comparison: Cohort C (4 Capsules b.i.d.): TIP/PBO vs Pooled PBO; Cohort C (4 capsules b.i.d.): TIP/PBO, Pooled PBO; Test type: Other; Odds Ratio, log = 3.41, 95% CI 2-sided [0.47 to 25.03] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 6: Comparison: Pooled TIP vs Pooled PBO; Test type: Other; Odds Ratio, log = 2.74, 95% CI 2-sided [0.47 to 16.07] — [estimate comment as in outcome 14, analysis 1]

15. Secondary Outcome: Time to First Hospitalization Due to Serious Respiratory-related Adverse Events
Description: Time to first hospitalization due to serious respiratory-related AEs was analyzed to define severity of pulmonary exacerbations compared to placebo. Participants were censored at the time of last contact if they did not have a hospitalization due to serious respiratory-related adverse events over the entire study period.
Time Frame: Baseline (Visit 101/Day 1) to Visit 202 (Day 169)
Population: Full Analysis Set
Measure: Median (95% Confidence Interval); unit: Day
Arm/Group | Cohort A (3 Capsules o.d.): TIP | Cohort A (3 Capsules o.d.): TIP/PBO | Cohort B (5 Capsules o.d.): TIP | Cohort B (5 Capsules o.d.): TIP/PBO | Cohort C (4 Capsules b.i.d.): TIP | Cohort C (4 Capsules b.i.d.): TIP/PBO | Pooled TIP | Pooled TIP/PBO | Pooled PBO
Number analyzed (Participants) | 14 | 13 | 15 | 14 | 15 | 15 | 44 | 42 | 21
Day | NA [93.00 to NA] — NA: Not estimable due to insufficient number of participants with events | NA [NA to NA] — NA: Not estimable due to insufficient number of participants with events | NA [60.00 to NA] — NA: Not estimable due to insufficient number of participants with events | NA [NA to NA] — NA: Not estimable due to insufficient number of participants with events | NA [NA to NA] — NA: Not estimable due to insufficient number of participants with events | NA [65.00 to NA] — NA: Not estimable due to insufficient number of participants with events | NA [NA to NA] — NA: Not estimable due to insufficient number of participants with events | NA [NA to NA] — NA: Not estimable due to insufficient number of participants with events | NA [NA to NA] — NA: Not estimable due to insufficient number of participants with events
Statistical Analysis 1: Comparison: Cohort A (3 Capsules o.d.): TIP vs Pooled PBO; Cohort A (3 capsules o.d.): TIP, Pooled PBO; Test type: Other; Hazard Ratio (HR) = 4.50, 95% CI 2-sided [0.77 to 26.42] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Cohort B (5 Capsules o.d.): TIP vs Pooled PBO; Cohort B (5 capsules o.d.): TIP, Pooled PBO; Test type: Other; Hazard Ratio (HR) = 2.00, 95% CI 2-sided [0.28 to 14.47] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Cohort B (5 Capsules o.d.): TIP/PBO vs Pooled PBO; Cohort B (5 capsules o.d.): TIP/PBO, Pooled PBO; Test type: Other; Hazard Ratio (HR) = 1.54, 95% CI 2-sided [0.20 to 11.60] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 4: Comparison: Cohort C (4 Capsules b.i.d.): TIP vs Pooled PBO; Cohort C (4 capsules b.i.d.): TIP, Pooled PBO; Test type: Other; Hazard Ratio (HR) = 0.67, 95% CI 2-sided [0.06 to 7.49] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 5: Comparison: Cohort C (4 Capsules b.i.d.): TIP/PBO vs Pooled PBO; Cohort C (4 capsules b.i.d.): TIP/PBO, Pooled PBO; Test type: Other; Hazard Ratio (HR) = 3.81, 95% CI 2-sided [0.62 to 23.29] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 6: Comparison: Pooled TIP vs Pooled PBO; Pooled TIP, Pooled PBO; Test type: Other; Hazard Ratio (HR) = 1.82, 95% CI 2-sided [0.35 to 9.45] — [estimate comment as in outcome 3, analysis 1]

16. Secondary Outcome: Serum Tobramycin Concentration
Description: The serum pharmacokinetic (PK) properties of tobramycin were assessed by evaluating tobramycin concentrations in serum collected from the non-cystic fibrosis bronchiectasis population post administration of o.d. or b.i.d. doses of TIP. Serum specimens for PK tobramycin concentration were assessed at Visit 101 (Day 1/start of treatment) 0 to 1 and 1 to 2 hours post-dose and Visit 102 (Day 8) 0 to 1 and 1 to 2 hours post-dose. Prior to protocol amendment #2, PK samples were assessed on Visits 103 (Day 29) rather than Visit 102. Only descriptive analysis performed.
Time Frame: Baseline (Visit 101/Day 1), Visit 102 (Day 8) and Visits 103 (Day 29): 0-1 hours and 1-2 hours post-dose.
Population: Pharmacokinetic Analysis Set. Prior to protocol amendment #2, PK samples were assessed on Visit 103 (Day 29) rather than Visit 102 (Day 8).
Measure: Mean (Standard Deviation); unit: microgram/milliliter
Arm/Group | Cohort A (3 Capsules o.d.): TIP | Cohort A (3 Capsules o.d.): TIP/PBO | Cohort B (5 Capsules o.d.): TIP | Cohort B (5 Capsules o.d.): TIP/PBO | Cohort C (4 Capsules b.i.d.): TIP | Cohort C (4 Capsules b.i.d.): TIP/PBO
Number analyzed (Participants) | 14 | 13 | 15 | 14 | 15 | 15
microgram/milliliter
  Visit 101 (Day 1)/0-1 hr post dose: number analyzed (Participants) | 12 | 11 | 11 | 11 | 14 | 11
  Visit 101 (Day 1)/0-1 hr post dose | 0.256 (0.144) | 0.479 (0.47) | 0.4 (0.259) | 0.441 (0.273) | 0.59 (0.37) | 0.321 (0.21)
  Visit 101 (Day 1)/1-2 hr post dose: number analyzed (Participants) | 11 | 11 | 11 | 11 | 13 | 10
  Visit 101 (Day 1)/1-2 hr post dose | 0.481 (0.287) | 0.571 (0.349) | 0.517 (0.392) | 0.624 (0.322) | 0.64 (0.338) | 0.476 (0.295)
  Visit 102 (Day 8)/0-1 hr post dose: number analyzed (Participants) | 0 | 1 | 1 | 1 | 1 | 2
  Visit 102 (Day 8)/0-1 hr post dose |  | 0 (NA) — NA: Not estimable due to insufficient number of participants with events | 1.81 (NA) — NA: Not estimable due to insufficient number of participants with events | 0.258 (NA) — NA: Not estimable due to insufficient number of participants with events | 1.4 (NA) — NA: Not estimable due to insufficient number of participants with events | 0.489 (0.257)
  Visit 102 (Day 8)/1-2 hr post dose: number analyzed (Participants) | 0 | 1 | 1 | 1 | 1 | 1
  Visit 102 (Day 8)/1-2 hr post dose |  | 0.18 (NA) — NA: Not estimable due to insufficient number of participants with events | 1.67 (NA) — NA: Not estimable due to insufficient number of participants with events | 0.588 (NA) — NA: Not estimable due to insufficient number of participants with events | 1.48 (NA) — NA: Not estimable due to insufficient number of participants with events | 0.447 (NA) — NA: Not estimable due to insufficient number of participants with events
  Visit 103 (Day 29)/0-1 hr post dose: number analyzed (Participants) | 9 | 11 | 8 | 9 | 9 | 7
  Visit 103 (Day 29)/0-1 hr post dose | 0.607 (0.455) | 0.0718 (0.0498) | 1.23 (1.08) | 0.103 (0.0983) | 1.05 (0.603) | 0.339 (0.274)
  Visit 103 (Day 29)/1-2 hr post dose: number analyzed (Participants) | 9 | 9 | 8 | 8 | 10 | 7
  Visit 103 (Day 29)/1-2 hr post dose | 0.768 (0.477) | 0.0818 (0.0972) | 1.37 (0.647) | 0.104 (0.096) | 1.05 (0.622) | 0.307 (0.24)

17. Secondary Outcome: Sputum Tobramycin Concentration
Description: The sputum pharmacokinetic (PK) properties of tobramycin were assessed by evaluating tobramycin concentrations in sputum collected from the non-cystic fibrosis bronchiectasis population post administration of o.d. or b.i.d. doses of TIP. Only descriptive analysis performed.
Time Frame: Baseline (Visit 101/Day 1): 0-1 hours and 1-2 hours post-dose; Visit 102 (Day 8):0-2 hours and 5-6 hours post-dose; Visits 103 (Day 29): 5 to 6 hours post-dose, Visit 104 (Day 57) and Visit 105 (Day 85): 3-4 hours post-dose.
Population: Pharmacokinetic Analysis Set. Prior to protocol amendment #2, Sputum specimens for PK assessments were collected at Visit 103 (Day 29) 5 to 6 hours rather than Visit 102 (Day 8) 0 to 2 and 5 to 6 hours and on Visit 105 (Day 85) 3 to 4 hours rather than Visit 104 (Day 57) 3 to 4 hours.
Measure: Mean (Standard Deviation); unit: microgram/milliliter
Arm/Group | Cohort A (3 Capsules o.d.): TIP | Cohort A (3 Capsules o.d.): TIP/PBO | Cohort B (5 Capsules o.d.): TIP | Cohort B (5 Capsules o.d.): TIP/PBO | Cohort C (4 Capsules b.i.d.): TIP | Cohort C (4 Capsules b.i.d.): TIP/PBO
Number analyzed (Participants) | 14 | 13 | 15 | 14 | 15 | 15
microgram/milliliter
  Visit 101 (Day 1)/0-1 hr post dose: number analyzed (Participants) | 13 | 11 | 10 | 12 | 13 | 11
  Visit 101 (Day 1)/0-1 hr post dose | 1750 (2160) | 637 (608) | 2640 (2680) | 2020 (2360) | 2820 (2250) | 2060 (1840)
  Visit 101 (Day 1)/1-2 hr post dose: number analyzed (Participants) | 14 | 11 | 8 | 11 | 10 | 7
  Visit 101 (Day 1)/1-2 hr post dose | 1100 (2480) | 204 (445) | 1650 (2340) | 1100 (2310) | 631 (441) | 610 (463)
  Visit 102 (Day 8)/0-2 hr post dose: number analyzed (Participants) | 14 | 9 | 7 | 11 | 11 | 9
  Visit 102 (Day 8)/0-2 hr post dose | 1440 (1470) | 2390 (2730) | 2460 (761) | 4290 (3730) | 1980 (2060) | 2290 (1560)
  Visit 102 (Day 8)/5-6 hr post dose: number analyzed (Participants) | 0 | 1 | 0 | 1 | 0 | 2
  Visit 102 (Day 8)/5-6 hr post dose |  | 32.4 (NA) — NA: Not estimable due to insufficient number of participants with events |  | 4460 (NA) — NA: Not estimable due to insufficient number of participants with events |  | 1200 (51.6)
  Visit 103 (Day 29)/5-6 hr post dose: number analyzed (Participants) | 9 | 7 | 6 | 7 | 4 | 7
  Visit 103 (Day 29)/5-6 hr post dose | 389 (554) | 136 (258) | 915 (1450) | 16.3 (28.6) | 620 (513) | 134 (175)
  Visit 104 (Day 57)/3-4 hr post dose: number analyzed (Participants) | 2 | 1 | 1 | 1 | 0 | 2
  Visit 104 (Day 57)/3-4 hr post dose | 198 (138) | 0 (NA) — NA: Not estimable due to insufficient number of participants with events | 96.4 (NA) — NA: Not estimable due to insufficient number of participants with events | 4540 (NA) — NA: Not estimable due to insufficient number of participants with events |  | 0 (0)
  Visit 105 (Day 85)/3-4 hr post dose: number analyzed (Participants) | 6 | 4 | 2 | 7 | 4 | 3
  Visit 105 (Day 85)/3-4 hr post dose | 791 (883) | 45.7 (75.8) | 101 (100) | 61 (108) | 2810 (2200) | 121 (166)

18. Secondary Outcome: Change From Baseline in Quality of Life Questionnaire for Bronchiectasis (QOL-B)-Physical Functioning
Description: The QoL-B consists of 37 items across 8 domains: Physical Functioning (PF), Role Functioning (RF), Vitality, Emotional Function (EF), Social Functioning (SF), Treatment Burden (TB), Health Perception (HP) and Respiratory Symptoms (RS). Each of the 37 items is scored from 1 to 4, and each of the 8 scale scores is standardized on a 0-100 point scale, with higher scores representing fewer symptoms or better functioning and HRQoL. A total score is not calculated since functioning can vary greatly from one domain to another. Only descriptive analysis performed.
Time Frame: Baseline, Visit 102 (Day 8), Visit 103 (Day 29), End of Treatment (Day 113) and Visit 202 (Day 169)
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Score on Scale
Arm/Group | Cohort A (3 Capsules o.d.): TIP | Cohort A (3 Capsules o.d.): TIP/PBO | Cohort B (5 Capsules o.d.): TIP | Cohort B (5 Capsules o.d.): TIP/PBO | Cohort C (4 Capsules b.i.d.): TIP | Cohort C (4 Capsules b.i.d.): TIP/PBO | Pooled TIP | Pooled TIP/PBO | Pooled PBO
Number analyzed (Participants) | 14 | 13 | 15 | 14 | 15 | 15 | 43 | 42 | 21
Score on Scale
  Baseline (BL): number analyzed (Participants) | 13 | 13 | 15 | 14 | 15 | 15 | 43 | 42 | 19
  Baseline (BL) | 51.33 (38.33) | 60.5 (28.60) | 45.8 (19.98) | 50.5 (33.04) | 46.2 (30.29) | 53.8 (26.72) | 47.6 (29.41) | 54.8 (29.10) | 49.8 (27.97)
  Change from BL at Day 8: number analyzed (Participants) | 13 | 12 | 12 | 14 | 15 | 15 | 40 | 41 | 19
  Change from BL at Day 8 | 5.6 (18.83) | -2.8 (14.35) | -6.7 (22.02) | -2.9 (18.06) | 0.9 (11.51) | 3.1 (14.44) | 0.2 (17.83) | -0.7 (15.62) | -7.4 (17.76)
  Change from BL at Day 29: number analyzed (Participants) | 13 | 12 | 10 | 13 | 15 | 14 | 38 | 39 | 19
  Change from BL at Day 29 | -2.1 (24.40) | -7.2 (16.44) | -5.3 (27.90) | -2.6 (8.41) | -0.4 (16.23) | -6.2 (27.48) | -2.3 (22.04) | -5.3 (19.05) | -1.1 (17.68)
  Change from BL at EoT: number analyzed (Participants) | 13 | 12 | 12 | 14 | 15 | 15 | 40 | 41 | 19
  Change from BL at EoT | -6.7 (18.66) | -6.1 (18.53) | -19.4 (23.00) | -6.7 (23.39) | -5.8 (31.36) | -9.8 (30.43) | -10.2 (25.44) | -7.6 (24.47) | 0.4 (20.30)
  Change from BL at Day 169: number analyzed (Participants) | 11 | 12 | 10 | 10 | 12 | 10 | 33 | 32 | 18
  Change from BL at Day 169 | 5.5 (25.27) | -3.3 (18.09) | 0.0 (22.44) | -1.3 (16.27) | -3.9 (26.43) | 7.3 (22.54) | 0.4 (24.43) | 0.6 (19.04) | -4.8 (16.77)

19. Secondary Outcome: Change From Baseline in Quality of Life Questionnaire for Bronchiectasis (QOL-B)-Role Functioning
Description: as for outcome 18
Time Frame: Baseline, Visit 102 (Day 8), Visit 103 (Day 29), End of Treatment (Day 113) and Visit 202 (Day 169)
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Score on Scale
Arm/Group | Cohort A (3 Capsules o.d.): TIP | Cohort A (3 Capsules o.d.): TIP/PBO | Cohort B (5 Capsules o.d.): TIP | Cohort B (5 Capsules o.d.): TIP/PBO | Cohort C (4 Capsules b.i.d.): TIP | Cohort C (4 Capsules b.i.d.): TIP/PBO | Pooled TIP | Pooled TIP/PBO | Pooled PBO
Number analyzed (Participants) | 14 | 13 | 15 | 14 | 15 | 15 | 43 | 42 | 21
Score on Scale
  Baseline (BL): number analyzed (Participants) | 13 | 13 | 15 | 14 | 15 | 15 | 43 | 42 | 19
  Baseline (BL) | 63.1 (24.28) | 67.2 (14.26) | 53.3 (21.68) | 64.3 (29.77) | 57.8 (26.86) | 67.6 (24.67) | 57.8 (24.11) | 66.3 (23.46) | 63.9 (19.79)
  Change from BL at Day 8: number analyzed (Participants) | 13 | 12 | 12 | 14 | 15 | 15 | 40 | 41 | 19
  Change from BL at Day 8 | 5.6 (14.36) | -2.2 (19.76) | 2.2 (20.17) | -1.4 (13.88) | 3.6 (17.43) | -4.2 (20.95) | 3.8 (17.01) | -2.7 (18.03) | -1.4 (14.67)
  Change from BL at Day 29: number analyzed (Participants) | 13 | 12 | 10 | 13 | 15 | 14 | 38 | 39 | 19
  Change from BL at Day 29 | 1.5 (19.66) | -1.1 (18.17) | 2.0 (21.33) | -1.0 (14.87) | -0.9 (19.82) | -4.5 (23.88) | 0.7 (19.65) | -2.3 (19.06) | 1.8 (16.00)
  Change from BL at EoT: number analyzed (Participants) | 13 | 12 | 12 | 14 | 15 | 15 | 40 | 41 | 19
  Change from BL at EoT | -0.5 (23.95) | -5.0 (24.47) | -0.4 (23.79) | -9.0 (25.30) | 0.9 (20.30) | -4.0 (24.27) | 0.0 (22.01) | -6.0 (24.17) | 1.0 (19.70)
  Change from BL at Day 169: number analyzed (Participants) | 11 | 12 | 10 | 10 | 12 | 10 | 33 | 32 | 18
  Change from BL at Day 169 | 10.3 (16.96) | -7.2 (17.17) | 10.7 (13.41) | -2.7 (21.82) | -6.1 (15.94) | 6.7 (16.92) | 4.4 (17.13) | -1.5 (18.99) | -4.4 (15.51)

20. Secondary Outcome: Change From Baseline in Quality of Life Questionnaire for Bronchiectasis (QOL-B)-Vitality
Description: as for outcome 18
Time Frame: Baseline, Visit 102 (Day 8), Visit 103 (Day 29), End of Treatment (Day 113) and Visit 202 (Day 169)
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Score on Scale
Arm/Group | Cohort A (3 Capsules o.d.): TIP | Cohort A (3 Capsules o.d.): TIP/PBO | Cohort B (5 Capsules o.d.): TIP | Cohort B (5 Capsules o.d.): TIP/PBO | Cohort C (4 Capsules b.i.d.): TIP | Cohort C (4 Capsules b.i.d.): TIP/PBO | Pooled TIP | Pooled TIP/PBO | Pooled PBO
Number analyzed (Participants) | 14 | 13 | 15 | 14 | 15 | 15 | 42 | 42 | 21
Score on Scale
  Baseline (BL): number analyzed (Participants) | 13 | 13 | 14 | 14 | 15 | 15 | 42 | 42 | 19
  Baseline (BL) | 56.4 (22.89) | 47.9 (17.21) | 52.4 (21.54) | 44.4 (26.51) | 47.4 (25.36) | 51.9 (18.63) | 51.9 (23.11) | 48.1 (20.92) | 46.2 (25.46)
  Change from BL at Day 8: number analyzed (Participants) | 13 | 12 | 11 | 14 | 15 | 15 | 39 | 41 | 19
  Change from BL at Day 8 | 6.8 (18.45) | 1.9 (24.54) | -6.1 (31.18) | 4.8 (17.27) | 5.2 (20.52) | 2.2 (11.27) | 2.6 (23.43) | 3.0 (17.57) | -2.9 (16.08)
  Change from BL at Day 29: number analyzed (Participants) | 13 | 12 | 9 | 13 | 15 | 14 | 37 | 39 | 19
  Change from BL at Day 29 | -4.3 (30.95) | 4.6 (15.23) | -9.9 (28.57) | 3.4 (18.36) | -0.7 (24.66) | -5.6 (23.77) | -4.2 (27.39) | 80.6 (19.74) | 1.8 (19.69)
  Change from BL at EoT: number analyzed (Participants) | 13 | 12 | 11 | 14 | 15 | 15 | 39 | 41 | 19
  Change from BL at EoT | -5.6 (25.26) | 2.8 (24.22) | -12.1 (26.04) | 3.2 (28.05) | -0.7 (29.24) | 2.2 (30.35) | -5.6 (26.77) | 2.7 (27.19) | -1.2 (23.97)
  Change from BL at Day 169: number analyzed (Participants) | 11 | 12 | 9 | 10 | 12 | 10 | 32 | 32 | 18
  Change from BL at Day 169 | 8.1 (20.55) | 3.7 (22.89) | 3.7 (24.22) | 2.2 (21.47) | -2.8 (22.78) | 1.1 (19.21) | 2.8 (22.22) | 2.4 (20.69) | -2.5 (20.36)

21. Secondary Outcome: Change From Baseline in Quality of Life Questionnaire for Bronchiectasis (QOL-B)-Emotional Functioning
Description: as for outcome 18
Time Frame: Baseline, Visit 102 (Day 8), Visit 103 (Day 29), End of Treatment (Day 113) and Visit 202 (Day 169)
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Score on Scale
Arm/Group | Cohort A (3 Capsules o.d.): TIP | Cohort A (3 Capsules o.d.): TIP/PBO | Cohort B (5 Capsules o.d.): TIP | Cohort B (5 Capsules o.d.): TIP/PBO | Cohort C (4 Capsules b.i.d.): TIP | Cohort C (4 Capsules b.i.d.): TIP/PBO | Pooled TIP | Pooled TIP/PBO | Pooled PBO
Number analyzed (Participants) | 14 | 13 | 15 | 14 | 15 | 15 | 42 | 42 | 21
Score on Scale
  Baseline (BL): number analyzed (Participants) | 13 | 13 | 14 | 14 | 15 | 15 | 42 | 42 | 18
  Baseline (BL) | 79.5 (14.28) | 71.2 (18.51) | 77.4 (17.73) | 74.4 (29.50) | 71.1 (18.86) | 76.1 (23.54) | 75.8 (17.15) | 74.0 (23.87) | 79.6 (16.96)
  Change from BL at Day 8: number analyzed (Participants) | 13 | 12 | 11 | 14 | 15 | 15 | 39 | 41 | 18
  Change from BL at Day 8 | 2.6 (11.48) | -4.2 (12.05) | -0.8 (13.67) | 2.4 (11.52) | 4.4 (18.33) | 4.4 (6.19) | 2.4 (14.80) | 1.2 (10.47) | -1.4 (11.87)
  Change from BL at Day 29: number analyzed (Participants) | 13 | 12 | 9 | 13 | 15 | 14 | 37 | 39 | 18
  Change from BL at Day 29 | 1.9 (11.36) | -4.9 (12.03) | 2.8 (13.18) | 3.8 (16.53) | 5.6 (13.24) | -1.2 (14.93) | 3.6 (12.35) | -0.6 (14.73) | -1.9 (12.31)
  Change from BL at EoT: number analyzed (Participants) | 13 | 12 | 11 | 14 | 15 | 15 | 39 | 41 | 18
  Change from BL at EoT | 1.3 (17.63) | -8.3 (22.19) | -9.1 (18.43) | 2.4 (32.26) | 1.1 (15.06) | -3.3 (14.36) | -1.7 (17.12) | -2.8 (23.76) | -2.3 (15.60)
  Change from BL at Day 169: number analyzed (Participants) | 11 | 12 | 9 | 10 | 12 | 10 | 32 | 32 | 17
  Change from BL at Day 169 | 6.1 (21.44) | -6.9 (15.00) | 7.4 (17.40) | 5.0 (18.51) | 0.0 (7.11) | 6.7 (21.45) | 4.2 (15.98) | 1.0 (18.78) | 3.9 (13.85)

22. Secondary Outcome: Change From Baseline in Quality of Life Questionnaire for Bronchiectasis (QOL-B)-Social Functioning
Description: as for outcome 18
Time Frame: Baseline, Visit 102 (Day 8), Visit 103 (Day 29), End of Treatment (Day 113) and Visit 202 (Day 169)
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Score on Scale
Arm/Group | Cohort A (3 Capsules o.d.): TIP | Cohort A (3 Capsules o.d.): TIP/PBO | Cohort B (5 Capsules o.d.): TIP | Cohort B (5 Capsules o.d.): TIP/PBO | Cohort C (4 Capsules b.i.d.): TIP | Cohort C (4 Capsules b.i.d.): TIP/PBO | Pooled TIP | Pooled TIP/PBO | Pooled PBO
Number analyzed (Participants) | 14 | 13 | 15 | 14 | 15 | 15 | 43 | 42 | 21
Score on Scale
  Baseline (BL): number analyzed (Participants) | 13 | 13 | 15 | 14 | 15 | 15 | 43 | 42 | 19
  Baseline (BL) | 66.2 (19.21) | 51.3 (22.53) | 36.5 (21.18) | 63.5 (26.17) | 48.5 (19.95) | 55.7 (26.80) | 49.7 (23.13) | 56.9 (25.22) | 51.9 (25.24)
  Change from BL at Day 8: number analyzed (Participants) | 13 | 12 | 12 | 14 | 15 | 15 | 40 | 41 | 19
  Change from BL at Day 8 | 3.0 (13.49) | 2.1 (23.61) | 29.6 (23.67) | -2.6 (12.49) | -0.7 (21.91) | 8.5 (15.66) | 9.6 (23.78) | 2.8 (17.67) | 5.0 (14.18)
  Change from BL at Day 29: number analyzed (Participants) | 13 | 12 | 10 | 13 | 15 | 14 | 38 | 39 | 19
  Change from BL at Day 29 | 4.9 (15.51) | -2.5 (26.05) | 22.8 (18.14) | -1.5 (24.50) | 2.6 (23.95) | 4.8 (19.89) | 8.7 (21.19) | 0.4 (23.07) | -1.2 (15.72)
  Change from BL at EoT: number analyzed (Participants) | 13 | 12 | 12 | 14 | 15 | 15 | 40 | 41 | 19
  Change from BL at EoT | 3.0 (21.71) | 2.1 (26.14) | 17.8 (27.89) | -5.6 (26.73) | 1.5 (30.10) | 5.7 (15.38) | 6.9 (27.25) | 0.8 (22.95) | -0.6 (18.04)
  Change from BL at Day 169: number analyzed (Participants) | 11 | 12 | 10 | 10 | 12 | 10 | 33 | 32 | 18
  Change from BL at Day 169 | 3.3 (24.27) | -5.1 (20.41) | 25.3 (21.73) | -4.2 (28.43) | -4.2 (25.42) | 11.9 (21.91) | 7.2 (26.36) | 0.5 (24.15) | -0.5 (19.37)

23. Secondary Outcome: Change From Baseline in Quality of Life Questionnaire for Bronchiectasis (QOL-B)-Treatment Burden
Description: as for outcome 18
Time Frame: Baseline, Visit 102 (Day 8), Visit 103 (Day 29), End of Treatment (Day 113) and Visit 202 (Day 169)
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Score on Scale
Arm/Group | Cohort A (3 Capsules o.d.): TIP | Cohort A (3 Capsules o.d.): TIP/PBO | Cohort B (5 Capsules o.d.): TIP | Cohort B (5 Capsules o.d.): TIP/PBO | Cohort C (4 Capsules b.i.d.): TIP | Cohort C (4 Capsules b.i.d.): TIP/PBO | Pooled TIP | Pooled TIP/PBO | Pooled PBO
Number analyzed (Participants) | 14 | 13 | 15 | 14 | 15 | 15 | 38 | 33 | 21
Score on Scale
  Baseline (BL): number analyzed (Participants) | 11 | 10 | 14 | 12 | 13 | 11 | 38 | 33 | 16
  Baseline (BL) | 67.7 (25.56) | 68.9 (26.09) | 64.3 (29.29) | 73.1 (18.63) | 56.4 (27.76) | 54.5 (27.42) | 62.6 (27.39) | 65.7 (24.75) | 64.6 (30.69)
  Change from BL at Day 8: number analyzed (Participants) | 10 | 9 | 11 | 12 | 13 | 11 | 34 | 32 | 13
  Change from BL at Day 8 | -2.2 (19.46) | -8.6 (29.28) | 0.0 (15.71) | -9.3 (17.62) | 4.3 (14.01) | 4.0 (7.49) | 1.0 (16.04) | -4.5 (19.73) | -2.6 (19.33)
  Change from BL at Day 29: number analyzed (Participants) | 11 | 8 | 8 | 10 | 12 | 9 | 31 | 27 | 13
  Change from BL at Day 29 | -9.1 (28.03) | -8.3 (27.70) | 8.3 (30.14) | -10.0 (22.50) | 1.9 (13.26) | -3.7 (25.46) | -0.4 (24.26) | -7.4 (24.27) | -5.1 (25.91)
  Change from BL at EoT: number analyzed (Participants) | 11 | 9 | 11 | 12 | 13 | 11 | 35 | 32 | 15
  Change from BL at EoT | -7.1 (21.81) | -8.6 (31.32) | -10.1 (16.07) | -14.8 (23.37) | 6.8 (26.66) | 1.0 (9.23) | -2.9 (22.92) | -7.6 (22.83) | -3.0 (30.13)
  Change from BL at Day 169: number analyzed (Participants) | 8 | 9 | 8 | 8 | 10 | 7 | 26 | 24 | 11
  Change from BL at Day 169 | 1.4 (26.19) | -3.7 (31.92) | 0.0 (13.28) | -4.2 (24.44) | 0.0 (17.37) | 12.7 (11.88) | 0.4 (18.72) | 0.9 (25.15) | -5.1 (18.16)

24. Secondary Outcome: Change From Baseline in Quality of Life Questionnaire for Bronchiectasis (QOL-B)-Health Perceptions
Description: as for outcome 18
Time Frame: Baseline, Visit 102 (Day 8), Visit 103 (Day 29), End of Treatment (Day 113) and Visit 202 (Day 169)
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Score on Scale
Arm/Group | Cohort A (3 Capsules o.d.): TIP | Cohort A (3 Capsules o.d.): TIP/PBO | Cohort B (5 Capsules o.d.): TIP | Cohort B (5 Capsules o.d.): TIP/PBO | Cohort C (4 Capsules b.i.d.): TIP | Cohort C (4 Capsules b.i.d.): TIP/PBO | Pooled TIP | Pooled TIP/PBO | Pooled PBO
Number analyzed (Participants) | 14 | 13 | 15 | 14 | 15 | 15 | 43 | 42 | 21
Score on Scale
  Baseline (BL): number analyzed (Participants) | 13 | 13 | 15 | 14 | 15 | 15 | 43 | 42 | 19
  Baseline (BL) | 41.0 (17.83) | 35.3 (19.29) | 33.1 (20.26) | 41.1 (27.83) | 39.4 (21.70) | 40.0 (20.70) | 37.7 (19.91) | 38.9 (22.52) | 41.7 (16.67)
  Change from BL at Day 8: number analyzed (Participants) | 13 | 12 | 12 | 14 | 15 | 15 | 40 | 41 | 19
  Change from BL at Day 8 | 7.1 (23.28) | 4.9 (20.24) | 10.0 (11.87) | -2.4 (13.25) | 5.6 (13.24) | 5.6 (15.96) | 7.4 (16.52) | 2.6 (16.50) | 0.0 (16.43)
  Change from BL at Day 29: number analyzed (Participants) | 13 | 12 | 10 | 13 | 15 | 14 | 38 | 39 | 19
  Change from BL at Day 29 | 7.1 (26.54) | 4.9 (20.24) | 12.8 (16.26) | 3.8 (19.73) | -1.1 (18.06) | -1.8 (26.19) | 5.3 (21.19) | 2.1 (22.02) | 3.1 (14.49)
  Change from BL at EoT: number analyzed (Participants) | 13 | 12 | 12 | 14 | 15 | 15 | 40 | 41 | 19
  Change from BL at EoT | -3.2 (25.35) | 0.7 (17.93) | -2.5 (15.28) | -3.6 (23.51) | 1.1 (23.12) | -0.6 (23.46) | -1.4 (21.43) | -1.2 (21.53) | 1.6 (16.67)
  Change from BL at Day 169: number analyzed (Participants) | 11 | 12 | 10 | 10 | 12 | 10 | 33 | 32 | 18
  Change from BL at Day 169 | 10.6 (13.99) | 0.0 (21.32) | 14.4 (19.72) | 6.7 (17.91) | -1.4 (11.70) | 9.2 (14.93) | 7.4 (16.30) | 4.9 (18.31) | 0.9 (19.57)

25. Secondary Outcome: Change From Baseline in Quality of Life Questionnaire for Bronchiectasis (QOL-B)-Respiratory Symptoms
Description: as for outcome 18
Time Frame: Baseline, Visit 102 (Day 8), Visit 103 (Day 29), End of Treatment (Day 113) and Visit 202 (Day 169)
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Score on Scale
Arm/Group | Cohort A (3 Capsules o.d.): TIP | Cohort A (3 Capsules o.d.): TIP/PBO | Cohort B (5 Capsules o.d.): TIP | Cohort B (5 Capsules o.d.): TIP/PBO | Cohort C (4 Capsules b.i.d.): TIP | Cohort C (4 Capsules b.i.d.): TIP/PBO | Pooled TIP | Pooled TIP/PBO | Pooled PBO
Number analyzed (Participants) | 14 | 13 | 15 | 14 | 15 | 15 | 43 | 42 | 21
Score on Scale
  Baseline (BL): number analyzed (Participants) | 13 | 13 | 15 | 14 | 15 | 15 | 43 | 42 | 19
  Baseline (BL) | 56.0 (13.05) | 53.8 (18.12) | 56.8 (17.63) | 55.9 (21.69) | 52.3 (22.39) | 61.9 (13.31) | 55.0 (17.98) | 57.4 (17.83) | 53.8 (14.42)
  Change from BL at Day 8: number analyzed (Participants) | 13 | 12 | 12 | 14 | 15 | 15 | 40 | 41 | 19
  Change from BL at Day 8 | 10.3 (6.83) | 6.5 (14.66) | 13.9 (16.12) | 3.3 (9.99) | 9.8 (12.30) | -0.6 (16.20) | 11.2 (12.05) | 2.8 (13.85) | 1.0 (12.09)
  Change from BL at Day 29: number analyzed (Participants) | 13 | 12 | 10 | 13 | 15 | 14 | 38 | 39 | 19
  Change from BL at Day 29 | 7.0 (11.94) | 0.6 (19.97) | 6.3 (24.57) | 3.6 (14.69) | 6.9 (22.57) | -5.7 (25.58) | 6.8 (19.65) | -0.7 (20.58) | 2.3 (13.48)
  Change from BL at EoT: number analyzed (Participants) | 13 | 12 | 12 | 14 | 15 | 15 | 40 | 41 | 19
  Change from BL at EoT | -0.4 (11.21) | 4.1 (15.65) | 1.9 (18.52) | -0.6 (20.73) | 6.7 (16.52) | -6.5 (26.18) | 2.9 (15.58) | -1.4 (21.59) | 4.0 (12.12)
  Change from BL at Day 169: number analyzed (Participants) | 11 | 12 | 10 | 10 | 12 | 10 | 33 | 32 | 18
  Change from BL at Day 169 | 7.1 (11.76) | 0.9 (16.42) | 10.7 (8.63) | -2.7 (24.33) | 5.6 (16.53) | 10.7 (12.52) | 7.6 (12.76) | 2.8 (18.57) | 1.6 (19.98)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study drug treatment until end of study treatment plus 30 days post treatment, up to a maximum duration of 134 days.
Description: Any sign or symptom that occurs during study treatment plus the 30 days post treatment.
Groups:
- Cohort C:4 Capsules b.i.d. TIP: Cohort C (4 capsules b.i.d.): Tobramycin inhalation powder (TIP)
Arm/Group | Cohort A (3 Capsules o.d.): TIP | Cohort A (3 Capsules o.d.): TIP/PBO | Cohort A (3 Capsules o.d.): PBO | Cohort B (5 Capsules o.d.): TIP | Cohort B (5 Capsules o.d.): TIP/PBO | Cohort B (5 Capsules o.d.): PBO | Cohort C:4 Capsules b.i.d. TIP | Cohort C (4 Capsules b.i.d.): TIP/PBO | Cohort C (4 Capsules b.i.d.): PBO
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/13 | 0/7 | 0/15 | 0/14 | 0/7 | 0/15 | 0/15 | 0/7
Serious Adverse Events (participants affected / at risk) | 4/14 | 2/13 | 0/7 | 4/15 | 3/14 | 2/7 | 2/15 | 4/15 | 1/7
Other Adverse Events (participants affected / at risk) | 12/14 | 12/13 | 6/7 | 10/15 | 10/14 | 7/7 | 13/15 | 14/15 | 5/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (3 Capsules o.d.): TIP (N=14) | Cohort A (3 Capsules o.d.): TIP/PBO (N=13) | Cohort A (3 Capsules o.d.): PBO (N=7) | Cohort B (5 Capsules o.d.): TIP (N=15) | Cohort B (5 Capsules o.d.): TIP/PBO (N=14) | Cohort B (5 Capsules o.d.): PBO (N=7) | Cohort C:4 Capsules b.i.d. TIP (N=15) | Cohort C (4 Capsules b.i.d.): TIP/PBO (N=15) | Cohort C (4 Capsules b.i.d.): PBO (N=7)
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bacterial disease carrier (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Infective exacerbation of bronchiectasis (Infections and infestations) | 3 | 0 | 0 | 2 | 1 | 0 | 0 | 3 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood creatinine abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Glomerular filtration rate decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (3 Capsules o.d.): TIP (N=14) | Cohort A (3 Capsules o.d.): TIP/PBO (N=13) | Cohort A (3 Capsules o.d.): PBO (N=7) | Cohort B (5 Capsules o.d.): TIP (N=15) | Cohort B (5 Capsules o.d.): TIP/PBO (N=14) | Cohort B (5 Capsules o.d.): PBO (N=7) | Cohort C:4 Capsules b.i.d. TIP (N=15) | Cohort C (4 Capsules b.i.d.): TIP/PBO (N=15) | Cohort C (4 Capsules b.i.d.): PBO (N=7)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cerumen impaction (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Deafness (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eustachian tube dysfunction (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Middle ear effusion (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1
Aerophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dental caries (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 3 | 2 | 1 | 1 | 0 | 2 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 2 | 1 | 1 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastric polyps (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lip swelling (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Oral pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia oral (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 0 | 0
Chest pain (General disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Discomfort (General disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Exercise tolerance decreased (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 1 | 2 | 0 | 1 | 3 | 2 | 2 | 0 | 1
Influenza like illness (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hepatotoxicity (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Food allergy (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Candida infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ear infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infective exacerbation of bronchiectasis (Infections and infestations) | 4 | 4 | 6 | 3 | 5 | 2 | 4 | 5 | 2
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Joint abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Labyrinthitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1 | 0 | 1 | 2 | 1 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1
Oral fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sputum purulent (Infections and infestations) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Viral infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Airway complication of anaesthesia (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypobarism (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 1 | 0 | 1 | 1 | 0 | 6 | 1 | 0
Blood electrolytes decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood urea increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 1 | 0 | 1 | 2 | 0 | 0 | 2 | 0 | 0
Eosinophil count abnormal (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Forced expiratory volume decreased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Forced vital capacity decreased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Glomerular filtration rate decreased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neutrophil count increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Protein urine present (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Sputum abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urine albumin/creatinine ratio increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urine protein/creatinine ratio increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Weight decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
White blood cell count increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Joint contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Muscle contracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ageusia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anosmia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 4 | 0 | 1 | 2 | 1 | 2 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasticity (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Calculus urinary (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Glycosuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Renal cyst (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 1 | 4 | 2 | 1 | 2 | 2 | 3
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1 | 3 | 2 | 2 | 4 | 2 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Dyspnoea paroxysmal nocturnal (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 2 | 3 | 0 | 2 | 1
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Increased viscosity of bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 2 | 1 | 2 | 0 | 1
Pulmonary pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory symptom (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1 | 0 | 1 | 0 | 0 | 3 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hot flush (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Novartis decided to close the recruitment of new subjects into this study earlier than scheduled. The early recruitment halt of the study was not due to safety or lack of efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-06-21): https://cdn.clinicaltrials.gov/large-docs/83/NCT02712983/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-21): https://cdn.clinicaltrials.gov/large-docs/83/NCT02712983/SAP_001.pdf